CLINICAL TRIAL: NCT04115839
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Filgotinib in Subjects With Active Psoriatic Arthritis Who Have an Inadequate Response or Are Intolerant to Biologic DMARD Therapy
Brief Title: Study to Evaluate the Efficacy and Safety of Filgotinib in Participants With Active Psoriatic Arthritis Who Have an Inadequate Response or Are Intolerant to Biologic DMARD Therapy
Acronym: PENGUIN 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-431-4567; 2019-002021-29 (EudraCT Number); JapicCTI-205201 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Filgotinib 200 mg (Main Study) (Experimental): Participants will receive filgotinib 200 mg + placebo to match (PTM) filgotinib 100 mg for up to 16 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Filgotinib 100 mg (Main Study) (Experimental): Participants will receive PTM filgotinib 200 mg + filgotinib 100 mg for up to 16 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Placebo (Main Study) (Placebo Comparator): Participants will receive PTM filgotinib 200 mg + PTM filgotinib 100 mg for up to 16 weeks.
  Interventions: Drug: Placebo to match filgotinib
- Filgotinib 200 mg (LTE) (Experimental): Participants will receive filgotinib 200 mg + PTM filgotinib 100 mg for up to 44 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Filgotinib 100 mg (LTE) (Experimental): Participants will receive PTM filgotinib 200 mg + filgotinib 100 mg for up to 44 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablets will be administered orally once daily with or without food.
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib 100 mg (LTE); Filgotinib 100 mg (Main Study); Filgotinib 200 mg (LTE); Filgotinib 200 mg (Main Study)
Drug: Placebo to match filgotinib — Tablets administered orally once daily with or without food.

SUMMARY:
The primary objective of this study is to evaluate the effect of filgotinib compared to placebo as assessed by the American College of Rheumatology 20% improvement (ACR20) response in participants with active psoriatic arthritis who have an inadequate response or are intolerant to biologic disease-modifying anti-rheumatic drugs (DMARD) therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participants who are 18-75 years of age (19-75 years of age at sites in Republic of Korea, 20-75 years of age at sites in Japan and Taiwan), on the day of signing initial informed consent
* Meet Classification Criteria for Psoriatic Arthritis (CASPAR)
* Have a history consistent with Psoriatic Arthritis (PsA) ≥ 6 months at Screening
* Have active PsA defined as ≥ 3 swollen joints (from a 66 swollen joint count [SJC]) and ≥ 3 tender joints (from a 68 tender joint count [TJC]) at Screening and Day 1; these may or may not be the same joints at Screening and Day 1
* Must have a documented history or active signs of at least one of the following at Screening

  * Plaque psoriasis
  * Nail changes attributed to psoriasis
* Have had inadequate response (lack of efficacy after ≥ 12 week duration of therapy) or intolerance to at least one and not more than 3 biologic DMARDs (bioDMARD) administered for the treatment of PsA or psoriasis, as per local guidelines / standard of care
* Prior to the first dose of study drug on Day 1, treatment with bioDMARD(s) should have been discontinued

Key Exclusion Criteria:

* Prior exposure to a janus kinase (JAK) inhibitor > 2 doses
* Any active / recent infection
* Any chronic and / or uncontrolled medical condition that would put the individual at increased risk during study participation or circumstances which may make a individual unlikely or unable to complete or comply with study procedures and requirements, per investigator judgement
* Any moderately to severely active musculoskeletal or skin disorder other than PsA or plaque psoriasis that would interfere with assessment of study parameters, as per judgement of investigator

NOTE: Prior history of reactive arthritis or axial spondyloarthritis is permitted if there is documentation of change in diagnosis to PsA or additional diagnosis of PsA

* Any history of an inflammatory arthropathy with onset before age of 16 years old
* Active autoimmune disease that would interfere with assessment of study parameters or increase risk to the individual by participating in the study, (e.g. uveitis, inflammatory bowel disease, uncontrolled thyroiditis, systemic vasculitis, transverse myelitis), per judgement of investigator
* Pregnancy or nursing females
* Active drug or alcohol abuse, as per judgement of investigator

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (59):
- United States (22):
  - Medvin Clinical Research, Covina, California
  - Omega Research Debary, LLC, DeBary, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Arthritis Center, Inc., Palm Harbor, Florida
  - Jefrey D. Lieberman, ND, P.C., Decatur, Georgia
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - St. Paul Rheumatology, P.A., Eagan, Minnesota
  - Arthritis Consultants, Inc., St Louis, Missouri
  - Atlantic Coast Research, Toms River, New Jersey
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Clinical Research Source Inc, Perrysburg, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Arthritis Group, PC, Philadelphia, Pennsylvania
  - PA Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - Articularis Healthcare Inc, dba, Columbia Arthritis Center, PA, Columbia, South Carolina
  - ACME Research, LLC, Orangeburg, South Carolina
  - Arthritis & Osteoporosis Clinic of Brazos Valley (Drug Shipment Address), College Station, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - West Virginia Research Institute PLLC, South Charleston, West Virginia
- Australia (3):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Rheumatology Research Unit, Maroochydore, Queensland
  - Emeritus Research, Camberwell, Victoria
- CHU UCL Namur - Site Godinne, Yvoir, Belgium
- G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec, Canada
- Czechia (2):
  - CCR Czech a.s., Pardubice
  - Reumatologie a Osteologie MEDICAL PLUS s.r.o., Rezidence Hradebni, Obchodni 1507, Uherske Hradiste, 68601, Uherské Hradiště
- Hungary (3):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Bekes Megeyi Kozponti Korhaz, Reumatologiai Osztaly, Gyula
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Mozgasszervi Rehabilitacios Osztaly, Szentes
- Japan (5):
  - Tokyo Medical University Hachioji Medical Center, Hachioji-shi
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - Daido Clinic, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Keio University Hospital, Tokyo
- Poland (8):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok, Podlaskie
  - NSZOZ Unica CR, Dabrówka
  - Centrum Badan Klinicznych PI-House sp. z o.o, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Centrum Medyczne AMED Warszawa Targowek, Warsaw
  - ARS RHEUMATICA Sp. Z.o.o., Warszawa, Mazowieckie
  - Centrum Medyczne Oporow, Wroclaw
- South Korea (3):
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - SMG - SNU Boramae Medical Center, Seoul
- Spain (7):
  - Hospital Universitario de Fuenlabrada - Rheumatology Department, Camino Del Molino no 2, Fuenlabrada, Madrid, 28942, Fuenlabrada
  - Hospital Universitario 12 de Octubre, Avenida de Cordoba, s/n, Madrid, Spain, 28041, Madrid
  - Hospital Universitario La Paz. Paseo de la Castellana 261, Madrid, 28046, Madrid
  - Corporacio Sanitaria Parc Tauli, Parc Tauli 1, Rheumatology Service, Sabadell, Barcelona, 08208, Sabadell
  - Hospital Universitario Marques de Valdecilla, Rheumatology Service, Avda. Valdecilla s/n, 39008, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Avenida Blasco Ibáñez, 17 Rheumatology Service, Valencia, Spain,, Valencia
- Taiwan (4):
  - Buddhist Dalin Tzu Chi Hospital, Dailin Township
  - Chi Mei Medical Center, Tainan
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Europe, Canada, Australia, and Asia. The first participant was screened on 13 November 2019. The last study visit occurred on 18 March 2021.
Pre-assignment Details: 170 participants were screened.
Groups:
- Filgotinib 200 mg (Main Study): Filgotinib 200 milligrams (mg) tablet orally once daily + placebo to match (PTM) filgotinib 100 mg tablet orally once daily for 16 weeks.
- Filgotinib 100 mg (Main Study): Filgotinib 100 mg tablet orally once daily + PTM filgotinib 200 mg tablet orally once daily for 16 weeks.
- Placebo (Main Study): PTM filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for 16 weeks.
- Filgotinib 200 mg From Filgotinib 200 mg (LTE): Long term extension (LTE):
  Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for up to 44.3 weeks. Participants received filgotinib 200 mg in the Main Study.
- Filgotinib 100 mg From Filgotinib 100 mg (LTE): Filgotinib 100 mg tablet orally once daily + PTM filgotinib 200 mg tablet orally once daily for up to 43.9 weeks. Participants received filgotinib 100 mg in the Main Study.
- Filgotinib 200 mg From Placebo (LTE): Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for up to 44.1 weeks. Participants received placebo in the Main Study.
- Filgotinib 100 mg From Placebo (LTE): Filgotinib 100 mg tablet orally once daily + PTM filgotinib 200 mg tablet orally once daily for up to 44 weeks. Participants received placebo in the Main Study.
Period: Main Study (Up to 16 Weeks)
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Started | 36 | 34 | 36 | 0 | 0 | 0 | 0
Completed | 18 | 20 | 18 | 0 | 0 | 0 | 0
Not Completed | 18 | 14 | 18 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 14 | 13 | 14 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 2 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: LTE Phase (After Week 16 to Week 63)
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Started | 0 (Participants who completed main study were randomised in LTE phase to receive filgotinib 200 mg or 100 mg.) | 0 (Participants who completed main study were randomised in LTE phase to receive filgotinib 200 mg or 100 mg.) | 0 (18 participants who completed main study did not enter LTE phase.) | 18 (Participants who completed main study were randomised in LTE phase to receive filgotinib 200 mg or 100 mg.) | 20 (Participants who completed main study were randomised in LTE phase to receive filgotinib 200 mg or 100 mg.) | 10 (10 participants who received placebo and completed main study were randomised in LTE phase to receive filgotinib 200 mg.) | 8 (8 participants who received placebo and completed main study were randomised in LTE phase to receive filgotinib 100 mg.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 18 | 20 | 10 | 8
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 17 | 19 | 10 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Filgotinib 200 mg (Main Study): Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study) | Total
Number analyzed (Participants) | 36 | 34 | 36 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10.5) | 54 (9.3) | 54 (10.5) | 55 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 18 | 45
  Male | 24 | 19 | 18 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 35 | 31 | 35 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 35 | 32 | 34 | 101
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 14 | 45
  Poland | 9 | 9 | 9 | 27
  Spain | 4 | 6 | 7 | 17
  Czechia | 2 | 2 | 2 | 6
  Canada | 2 | 1 | 0 | 3
  Australia | 1 | 0 | 1 | 2
  Hungary | 1 | 0 | 1 | 2
  Japan | 1 | 1 | 0 | 2
  South Korea | 0 | 0 | 1 | 1
  Taiwan | 0 | 0 | 1 | 1
Psoriatic Arthritis Disease Activity Score (PASDAS) [Mean (Standard Deviation); unit: score on a scale] — PASDAS is a composite disease activity measure for psoriatic arthritis. The score of PASDAS range from 0 -10, lower score indicates better function.
  score on a scale | 5.9 (0.97) | 5.7 (1.07) | 5.6 (0.93) | 5.7 (0.99)
Disease Activity in Psoriatic Arthritis (DAPSA) [Mean (Standard Deviation); unit: score on a scale] — DAPSA score is the sum of swollen joint count (66 joints), tender joint count (68 joints), CRP (mg/dL), patient's global assessment of PsA pain intensity (PGAPI) [using visual analogue scale (VAS) on a scale of 0-100, 0 = no pain and 100 = serious pain), and patient's global assessment of disease activity (PGADA) (using VAS on a scale of 0-100, 0 = very well and 10 = very poor). DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. Lower scores indicate better function.
  score on a scale | 45.9 (22.64) | 42.8 (22.05) | 43.1 (23.26) | 44.0 (22.49)
Physician's Global Assessment of Psoriasis (PhGAP) [Mean (Standard Deviation); unit: score on a scale] — The PhGAP is used to determine the participant's psoriasis lesions overall at a given time point. The participant's psoriasis disease activity is assessed by a physician according to the grades of induration, erythema and scaling on a scale of 0 to 5. The sum of the three grades will be used to obtain the total average score. PhGAP is based on the total average score on a scale of 0-5, where, 0=cleared, 1=minimal, 2=mild, 3=moderate, 4=marked and 5=severe. Lower scores indicates better function. Population: Participants in the FAS with ≥ 3% BSA at baseline were analyzed.
  score on a scale
    number analyzed (Participants) | 16 | 17 | 16 | 49
    (all) | 2.7 (0.79) | 2.8 (0.95) | 2.9 (0.81) | 2.8 (0.84)
Modified Nail Psoriasis Severity Index (mNAPSI) [Mean (Standard Deviation); unit: score on a scale] — mNAPSI is used to assess each nail abnormality for each of the participant's nails. Each finger has a score between 0 and 13. The total mNAPSI score is the sum of all abnormalities of individual score across all fingers, and the total mNAPSI score ranges from 0 to 130. Lower numbers indicate fewer nail abnormalities. Population: Participants in the FAS with Psoriatic Nail Involvement at Baseline were analyzed.
  score on a scale
    number analyzed (Participants) | 25 | 25 | 30 | 80
    (all) | 11 (9.7) | 15 (21.4) | 10 (7.1) | 12 (13.8)
Leeds Enthesitis Index (LEI) [Mean (Standard Deviation); unit: score on a scale] — Enthesitis is assessed using LEI. The enthesitis examination by LEI evaluated the presence or absence of pain by applying local pressure on 6 anatomical sites: medial femoral condyle (left and right), lateral epicondyle (left and right) and the achilles tendon insertion (left and right). Enthesitis at each site was scored as 0 = enthesitis absent and 1 = enthesitis present. The total score ranges from 0 to 6, higher scores indicates greater degree of enthesitis. Population: Participants in the FAS with enthesitis at baseline were analyzed.
  score on a scale
    number analyzed (Participants) | 22 | 22 | 24 | 68
    (all) | 2 (1.7) | 2 (1.6) | 1 (1.2) | 2 (1.5)
12-Item Psoriatic Arthritis Impact of Disease (PsAID-12) [Mean (Standard Deviation); unit: score on a scale] — The PsAID questionnaire assesses the impact of PsA on people's lives. The PsAID is calculated based on 12 numerical rating scales (NRS) questions. Each NRS is assessed as a number between 0 and 10. Total score is calculated as the sum of the individual scores, (some of which were multiplied by a weighting factor) divided by 20 for a total possible score of 0 to 10, where higher score indicates worse impact of disease.
  score on a scale | 5.2 (1.94) | 5.1 (2.33) | 4.8 (2.10) | 5.0 (2.11)
Tender Joint Count Based on 68 Joints (TJC68) [Mean (Standard Deviation); unit: tender joint count] — TJC68 is an assessment of 68 joints. Each joint was evaluated as 'normal', 'tender', 'tender and swollen' or 'not able to evaluate'. It is derived as the sum of all tender joints. The overall tender joint count ranged from 0 to 68, with a higher score indicating a greater degree of tenderness.
  tender joint count | 23 (17.2) | 21 (14.6) | 22 (15.3) | 22 (15.6)
Swollen Joint Count Based on 66 Joints (SJC66) [Mean (Standard Deviation); unit: swollen joint count] — SJC66 is an assessment of 66 joints. Each joint was evaluated as 'normal', 'swollen', 'tender and swollen' or 'not able to evaluate'. It is derived as the sum of all swollen joints. The overall swollen joint count ranged from 0 to 66, with a higher score indicating a greater degree of swelling.
  swollen joint count | 11 (6.7) | 10 (8.7) | 10 (8.9) | 10 (8.1)
Patient's Global Assessment of Disease Activity (PGADA) [Mean (Standard Deviation); unit: score on a scale] — PGADA is assessed by the participants using a VAS on a scale of 0 (very well) to 100 (very poor).
  score on a scale | 56 (22.4) | 55 (24.7) | 53 (21.1) | 55 (22.6)
Physician's Global Assessment of Disease Activity (PhGADA) [Mean (Standard Deviation); unit: score on a scale] — PhGADA is assessed by the physician using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity).
  score on a scale | 63 (13.8) | 63 (14.0) | 59 (14.5) | 62 (14.1)
Health Assessment Questionnaire Disability Index (HAQ-DI)'s Pain Assessment [Mean (Standard Deviation); unit: score on a scale] — Participants assessed their pain severity using a VAS on a scale of 0 (no pain) to 100 (severe pain).
  score on a scale | 61 (19.3) | 56 (23.3) | 57 (23.4) | 58 (21.9)
High-Sensitivity C- Reactive Protein (hsCRP) [Mean (Standard Deviation); unit: milligrams per liter (mg/L)] | 8.03 (18.347) | 7.58 (10.361) | 8.20 (12.707) | 7.94 (14.149)
Disease Activity Score 28 (DAS28) C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: score on a scale] — DAS28(CRP) is a measure of the participant's disease activity calculated using the tender joint count (28 joints), swollen joint count (28 joints), PGADA [using a VAS on a scale of 0 (very well) to 100 (very poor)] and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity.
  score on a scale | 4.8 (0.98) | 4.8 (0.97) | 4.8 (1.00) | 4.8 (0.97)
Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: score on a scale] — PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). A higher score indicates more severe disease. Population: Participants in the FAS with psoriasis covering >=3% of the BSA at baseline were analyzed.
  score on a scale
    number analyzed (Participants) | 16 | 17 | 16 | 49
    (all) | 8.5 (6.54) | 9.6 (6.43) | 9.1 (6.25) | 9.1 (6.29)
Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index [Mean (Standard Deviation); unit: score on a scale] — The enthesitis examination is based on the 16 anatomical sites. SPARCC enthesitis index has an overall total score ranging from 0 to 16. Higher score indicates a greater number of sites that are affected by enthesitis. Population: Participants in FAS with Enthesitis at Baseline were analyzed.
  score on a scale
    number analyzed (Participants) | 22 | 22 | 24 | 68
    (all) | 4 (3.8) | 6 (4.4) | 4 (2.8) | 5 (3.7)
Leeds Dactylitis Index (LDI) [Mean (Standard Deviation); unit: score on a scale] — LDI quantitatively measures dactylitis using the circumference of involved digits and control digits and tenderness of involved digits. LDI measures the ratio of the circumference of the affected digit to the circumference of the digit on the contralateral hand or foot using a Leeds Dactylometer. LDI score is calculated based on the circumference of the dactylitic finger/toe (mm), circumference of the contralateral digit (mm), tenderness score. Tenderness of affected digits is assessed on a scale from 0 [no tenderness] to 3 [tender and withdrawn]. A higher LDI indicates worse dactylitis. Population: Participants in FAS with Dactylitis at Baseline were analyzed.
  score on a scale
    number analyzed (Participants) | 15 | 6 | 9 | 30
    (all) | 54.8 (83.24) | 21.9 (26.26) | 22.1 (12.91) | 38.4 (61.55)
Tender Dactylitis Count (TDC) [Mean (Standard Deviation); unit: tender dactylitis count] — Tender score (0 = no tenderness, 1 = tender, 2 = tender and wince, 3 = tender and withdraw) is collected for Dactylitis Assessments on the Dactylitis Score Sheet that was used for calculation of LDI total score. Tender dactylitis count (TDC) equals the number of tender fingers and toes (tendor score >0). For participants with dactylitis status absent for all the fingers and toes, the TDC will be set as 0. The total score range of TDC is from 0 to 60, higher scores indicate greater presence of dactylitis. Population: Participants in the FAS with dactylitis at baseline were analyzed.
  tender dactylitis count
    number analyzed (Participants) | 15 | 6 | 9 | 30
    (all) | 3 (4.9) | 1 (0.6) | 1 (0.9) | 2 (3.6)
Health Assessment Questionnaire-Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: score on a scale] — The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). When 6 or more categories are non-missing, total possible score is 3. If more than 2 categories are missing, the HAQ-DI score is set to missing.
  score on a scale | 1.24 (0.637) | 1.03 (0.612) | 1.13 (0.557) | 1.14 (0.603)
Functional Assessment of Chronic Illness Therapy (FACIT)- Fatigue [Mean (Standard Deviation); unit: score on a scale] — FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 0 to 52. Higher scores indicate less fatigue.
  score on a scale | 25.9 (12.98) | 30.9 (10.08) | 31.0 (10.66) | 29.2 (11.48)
36-item Short-Form Version 2 (SF-36v2) [Mean (Standard Deviation); unit: score on a scale] — The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (MCS and PCS). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning.
  score on a scale
    Mental Component Summary (MCS) | 45.8 (11.97) | 48.1 (8.79) | 49.8 (12.20) | 47.9 (11.15)
    Physical Component Summary (PCS) | 33.7 (8.13) | 35.5 (9.41) | 35.7 (9.05) | 34.9 (8.83)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20% Improvement Response at Week 12
Description: ACR20 response is achieved when the participant has: ≥ 20% improvement (reduction) from baseline in tender joint count based on 68 joints (TJC68), swollen joint count based on 66 joints (SJC66) and in at least 3 of the following 5 items: patient's global assessment of disease activity (PGADA) using a visual analogue scale (VAS) on a scale of 0 (very well) to 100 (very poor); physician's global assessment of disease activity (PHGADA) using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity); health assessment questionnaire-disability index (HAQ-DI) inclusive of activities scored on a scale of 0 (no disability) to 3 (completely disabled); HAQ-DI pain assessment using VAS on a scale of 0 (no pain) to 100 (serious pain), and high-sensitivity C-reactive protein (hsCRP).
Time Frame: Week 12
Population: Full Analysis Set (FAS) included all randomized participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants | 60.0 [43.5 to 76.5] | 35.3 [17.8 to 52.8] | 33.1 [17.0 to 49.1]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.022, Multiple imputation method — The stratification factors (Geographic Region, Concurrent Use of conventional synthetic (cs) DMARD(s) and/or Apremilast at Randomization, Prior Use of biologic (bio)DMARD(s)) and treatment groups were included in the imputation model as covariates; Difference in response rates = 26.9, 95% CI 2-sided [4.3 to 49.6]
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.89, Multiple imputation method — The stratification factors (Geographic Region, Concurrent Use of csDMARD(s) and/or Apremilast at Randomization, Prior Use of bioDMARD(s)) and treatment groups were included in the imputation model as covariates; Difference in response rates = 2.2, 95% CI 2-sided [-20.5 to 25.0]

2. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) at Weeks 4 and 16
Description: PASDAS is a composite disease activity measure for psoriatic arthritis. The PASDAS includes the following components: PGADA [using a VAS on a scale of 0 (very well) to 100 (very poor)]; PhGADA [using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity)]; 36-item short form survey (SF-36) [a questionnaire which measures quality of life across eight domains used to determine a physical component summary (PCS) with a score range of 0-100, higher scores indicates better health status]; TJC68; SJC66; leeds enthesitis index (LEI) [assessed at 6 sites with a score range of 0 to 6, higher scores indicates higher degree of enthesitis]; Tender dactylitis count (TDC) [with a score range of 0 to 60, higher score indicates higher degree of dactylitis]; C-reactive protein (CRP). The score of PASDAS ranges from 0-10, lower scores indicates better function. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 35
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 34 | 33 | 34
  Change from Baseline at Week 4 | -1.2 (1.34) | -0.8 (0.73) | -0.6 (0.96)
  Change from Baseline at Week 16: number analyzed (Participants) | 31 | 33 | 32
  Change from Baseline at Week 16 | -2.1 (1.73) | -1.4 (1.19) | -0.9 (1.08)

3. Secondary Outcome: Change From Baseline in PASDAS at Week 48
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Filgotinib 200 mg From Filgotinib 200 mg (LTE): Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for up to 44.3 weeks. Participants received filgotinib 200 mg in the Main Study.
- Filgotinib 100 mg From Filgotinib 100 mg (LTE): Filgotinib 100 mg tablet orally once daily+ PTM filgotinib 200 mg tablet orally once daily for up to 43.9 weeks. Participants received filgotinib 100 mg in the Main Study.
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 8 | 9 | 4 | 3
score on a scale | -3.3 (1.69) | -2.0 (1.35) | -1.7 (0.57) | 0.0 (0.30)

4. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) Response at Weeks 4, 8, 12, and 16
Description: MDA is a measure to indicate disease remission, and is based on a composite score of 7 domains. A participant is considered as having achieved the MDA if the participant fulfills at least 5 of the following 7 criteria: TJC68 ≤1; SJC66 ≤1; Psoriatic arthritis disease activity score (PASI) ≤1 for participants with psoriasis covering BSA <3% [PASI evaluates the severity and extent of psoriasis. In PASI, body is divided into four parts, head and neck, upper limb, trunk and lower limbs. Each area is assessed for erythema, induration and scaling, each rated on a scale of 0 to 4. The total score ranges from 0 (no disease) to 72 (maximal disease)]; PGAPI ≤15 [using VAS on a scale of 0 (no pain) to 100 (serious pain)]; PGADA ≤20 [using VAS on a scale of 0 (very well) to 100 (very poor)]; HAQ-DI score ≤0.5; LEI score ≤1 for participants with enthesitis at baseline.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 4: number analyzed (Participants) | 36 | 34 | 35
  Week 4 | 5.6 [0.0 to 14.4] | 8.8 [0.0 to 19.8] | 11.4 [0.0 to 23.4]
  Week 8: number analyzed (Participants) | 32 | 34 | 34
  Week 8 | 15.6 [1.5 to 29.8] | 11.8 [0.0 to 24.1] | 14.7 [1.3 to 28.1]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 21.2 [5.7 to 36.7] | 17.6 [3.4 to 31.9] | 8.8 [0.0 to 19.8]
  Week 16: number analyzed (Participants) | 32 | 33 | 33
  Week 16 | 34.4 [16.4 to 52.4] | 24.2 [8.1 to 40.4] | 12.1 [0.0 to 24.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.39, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors (geographic Region, concurrent Use of csDMARD(s) and/or Apremilast at Randomization, prior use of bioDMARD(s)) in the model; Difference in response rates = -5.9, 95% CI 2-sided [-21.6 to 9.9] — 95% confidence interval (CI) for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.65, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -2.6, 95% CI 2-sided [-19.7 to 14.5] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.86, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 0.9, -19.4% CI 2-sided [-19.4 to 21.3] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.70, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -2.9, 95% CI 2-sided [-22.0 to 16.1] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.15, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 12.4, 95% CI 2-sided [-7.5 to 32.3] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.30, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 8.8, 95% CI 2-sided [-10.1 to 27.7] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.035, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 22.3, 95% CI 2-sided [-0.7 to 45.2] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.22, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 12.1, 95% CI 2-sided [-9.3 to 33.5] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Achieved MDA Response at Weeks 20, 24, 28, 36, and 48
Description: as for outcome 4
Time Frame: Weeks 20, 24, 28, 36, and 48
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Week 20 | 30.8 [1.8 to 59.7] | 21.1 [0.1 to 42.0] | 40.0 [4.6 to 75.4] | 0 [0.0 to 6.3]
  Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Week 24 | 38.5 [8.2 to 68.8] | 43.8 [16.3 to 71.2] | 71.4 [30.8 to 100.0] | 28.6 [0.0 to 69.2]
  Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Week 28 | 37.5 [0.0 to 77.3] | 36.4 [3.4 to 69.3] | 50.0 [0.0 to 100.0] | 20.0 [0.0 to 65.1]
  Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Week 36 | 55.6 [17.5 to 93.6] | 30.0 [0.0 to 63.4] | 50.0 [0.0 to 100.0] | 20.0 [0.0 to 65.1]
  Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Week 48 | 62.5 [22.7 to 100.0] | 11.1 [0.0 to 37.2] | 75.0 [20.1 to 100.0] | 0 [0.0 to 16.7]

6. Secondary Outcome: Percentage of Participants Who Achieved Very Low Disease Activity (VLDA) Response at Weeks 4, 8, 12, and 16
Description: VLDA is a measure to indicate disease remission, and is based on a composite score of 7 domains. A participant is considered as having achieved the VLDA if the participant fulfills all the seven criteria: TJC68 ≤1; SJC66 ≤1; PASI score ≤1 for participants with psoriasis covering BSA <3% [PASI evaluates the severity and extent of psoriasis. In PASI, body is divided into four parts, head and neck, upper limb, trunk and lower limbs. Each area is assessed for erythema, induration and scaling, each rated on a scale of 0 to 4. The total score ranges from 0 (no disease) to 72 (maximal disease)]; PGAPI ≤15 [using VAS on a scale of 0 (no pain) to (serious pain)]; PGADA ≤20 [using VAS on a scale of 0 (very well) to 100 (very poor)]; HAQ-DI score ≤0.5; LEI score ≤1 with participants with enthesitis at baseline.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Filgotinib 200 mg (Main Study): Filgotinib 200 mg tablet orally once daily+ PTM filgotinib 100 mg tablet orally once daily for 16 weeks.
- Placebo (Main Study): PTM filgotinib 200 mg tablet orally once daily+ PTM filgotinib 100 mg tablet orally once daily for 16 weeks.
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 4: number analyzed (Participants) | 36 | 34 | 35
  Week 4 | 0 [0.0 to 1.4] | 0 [0.0 to 1.5] | 0 [0.0 to 1.4]
  Week 8: number analyzed (Participants) | 32 | 34 | 34
  Week 8 | 3.1 [0.0 to 10.7] | 0 [0.0 to 1.5] | 0 [0.0 to 1.5]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 3.0 [0.0 to 10.4] | 5.9 [0.0 to 15.3] | 0 [0.0 to 1.5]
  Week 16: number analyzed (Participants) | 32 | 33 | 33
  Week 16 | 3.1 [0.0 to 10.7] | 6.1 [0.0 to 15.7] | 3.0 [0.0 to 10.4]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-2.8 to 2.8] — 95% CI for response rate and difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-2.9 to 2.9] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 3.1, 95% CI 2-sided [-5.9 to 12.2] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-2.9 to 2.9] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 3.0, 95% CI 2-sided [-5.8 to 11.9] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 5.9, 95% CI 2-sided [-5.0 to 16.7] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 0.1, 95% CI 2-sided [-11.4 to 11.6] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 3.0, 95% CI 2-sided [-10.0 to 16.1] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Percentage of Participants Who Achieved VLDA Response at Weeks 20, 24, 28, 36, and 48
Description: as for outcome 6
Time Frame: Weeks 20, 24, 28, 36, and 48
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Week 20 | 7.7 [0.0 to 26.0] | 0 [0.0 to 2.6] | 10.0 [0.0 to 33.6] | 0 [0.0 to 6.3]
  Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Week 24 | 7.7 [0.0 to 26.0] | 12.5 [0.0 to 31.8] | 14.3 [0.0 to 47.4] | 0 [0.0 to 7.1]
  Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Week 28 | 12.5 [0.0 to 41.7] | 0 [0.0 to 4.5] | 0 [0.0 to 12.5] | 0 [0.0 to 10.0]
  Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Week 36 | 22.2 [0.0 to 54.9] | 10.0 [0.0 to 33.6] | 0 [0.0 to 12.5] | 0 [0.0 to 10.0]
  Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Week 48 | 0 [0.0 to 6.3] | 0 [0.0 to 5.6] | 0 [0.0 to 12.5] | 0 [0.0 to 16.7]

8. Secondary Outcome: Change From Baseline in Disease Activity in Psoriatic Arthritis (DAPSA) at Weeks 2, 4, 8, 12, and 16
Description: DAPSA is calculated by summing the following components: TJC68; SJC66; PGADA [using VAS on a scale of 0 (very well) to 100 very poor)]; PGAPI [using a VAS on a scale of 0 (no pain) to 100 (serious pain)] and CRP. DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Filgotinib 100 mg (Main Study): Filgotinib 100 mg tablet orally once daily+ PTM filgotinib 200 mg tablet orally once daily for 16 weeks.
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 33 | 35
  Change from Baseline at Week 2 | -11.6 (19.12) | -9.4 (14.11) | -2.9 (16.01)
  Change from Baseline at Week 4: number analyzed (Participants) | 35 | 34 | 34
  Change from Baseline at Week 4 | -15.1 (18.48) | -11.5 (12.53) | -8.0 (19.32)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 33
  Change from Baseline at Week 8 | -22.0 (21.73) | -14.4 (14.96) | -14.4 (20.15)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 33
  Change from Baseline at Week 12 | -25.2 (24.43) | -15.8 (19.32) | -14.9 (16.43)
  Change from Baseline at Week 16: number analyzed (Participants) | 31 | 33 | 32
  Change from Baseline at Week 16 | -26.3 (23.48) | -19.4 (18.13) | -16.6 (15.61)

9. Secondary Outcome: Change From Baseline in DAPSA at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 8
Time Frame: Baseline, 18, 20, 24, 28, 36, 48, and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
score on a scale
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -27.0 (22.87) | -23.5 (18.80) | -9.3 (9.10) | -5.3 (9.72)
  Change from Baseline at Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Change from Baseline at Week 20 | -32.1 (29.72) | -20.5 (15.12) | -9.6 (11.79) | 1.1 (16.48)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Change from Baseline at Week 24 | -28.8 (37.40) | -22.1 (18.37) | -6.9 (6.51) | -5.4 (15.02)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 4
  Change from Baseline at Week 28 | -37.3 (26.49) | -24.1 (20.79) | -3.0 (7.61) | -5.3 (20.48)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -44.9 (27.81) | -23.6 (18.30) | -1.3 (10.75) | -9.9 (13.51)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -40.5 (31.97) | -28.5 (20.68) | -16.3 (21.00) | -2.3 (17.56)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | -86.2 (NA) — Standard deviation (SD) cannot be calculated for 1 participant. | -18.5 (NA) — Standard deviation (SD) cannot be calculated for 1 participant. | -12.9 (11.80) | 1.8 (23.75)

10. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Psoriasis (PhGAP) at Weeks 2, 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the Body Surface Area (BSA) at Baseline
Description: The PhGAP is used to determine the participant's psoriasis lesions overall at a given time point. The participant's psoriasis disease activity is assessed by a physician according to the grades of induration, erythema, and scaling on a scale of 0 to 5. The sum of the three grades is used to obtain the total average score. PhGAP is based on the total average score on a scale of 0-5 where, 0 = cleared, 1 = minimal, 2 = mild, 3 = moderate, 4 = marked, and 5 = severe. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with psoriasis covering >=3% of the BSA at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 16 | 17 | 16
score on a scale
  Change from Baseline at Week 2 | -1 (0.9) | 0 (0.7) | 0 (0.9)
  Change from Baseline at Week 4: number analyzed (Participants) | 16 | 17 | 15
  Change from Baseline at Week 4 | -1 (1.1) | 0 (0.7) | 0 (1.1)
  Change from Baseline at Week 8: number analyzed (Participants) | 16 | 17 | 14
  Change from Baseline at Week 8 | -1 (0.9) | 0 (0.8) | -1 (1.1)
  Change from Baseline at Week 12: number analyzed (Participants) | 16 | 17 | 13
  Change from Baseline at Week 12 | -1 (1.0) | -1 (0.7) | -1 (0.8)
  Change from Baseline at Week 16: number analyzed (Participants) | 15 | 17 | 14
  Change from Baseline at Week 16 | -2 (1.0) | 0 (0.7) | 0 (0.9)

11. Secondary Outcome: Change From Baseline in PhGAP at Weeks 18, 20, 24, 28, 36, and 48 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: as for outcome 10
Time Frame: Baseline, 18, 20, 24, 28, 36, and 48 weeks
Population: Participants in the FAS with psoriasis covering >=3% of the BSA at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 16 | 17 | 5 | 2
score on a scale
  Change from Baseline at Week 18: number analyzed (Participants) | 7 | 7 | 3 | 2
  Change from Baseline at Week 18 | -2 (1.4) | -1 (0.5) | -1 (0.6) | 0 (0.0)
  Change from Baseline at Week 20: number analyzed (Participants) | 6 | 8 | 5 | 2
  Change from Baseline at Week 20 | -1 (0.9) | 0 (0.9) | -1 (0.8) | 0 (0.0)
  Change from Baseline at Week 24: number analyzed (Participants) | 7 | 7 | 4 | 2
  Change from Baseline at Week 24 | -2 (1.1) | 0 (0.5) | -2 (0.8) | -1 (0.7)
  Change from Baseline at Week 28: number analyzed (Participants) | 3 | 6 | 3 | 1
  Change from Baseline at Week 28 | -1 (0.6) | -1 (0.4) | -1 (1.2) | -1 (NA) — SD cannot be calculated for 1 participant.
  Change from Baseline at Week 36: number analyzed (Participants) | 4 | 5 | 4 | 1
  Change from Baseline at Week 36 | -2 (0.6) | 0 (0.5) | -1 (0.8) | 0 (NA) — SD cannot be calculated for 1 participant.
  Change from Baseline at Week 48: number analyzed (Participants) | 4 | 5 | 4 | 1
  Change from Baseline at Week 48 | -1 (1.0) | 0 (0.4) | -1 (0.8) | 0 (NA) — SD cannot be calculated for 1 participant.

12. Secondary Outcome: Change From Baseline in Modified Nail Psoriasis Severity Index (mNAPSI) at Weeks 4, 8, 12, and 16 in Participants With Psoriatic Nail Involvement at Baseline
Description: mNAPSI is used to assess each nail abnormality for each of the participant's nails. Three features or groups of features (pitting, onycholysis together with oil-drop dyschromia, and crumbling) of each fingernail are graded on a scale from 0 (no onycholysis together with oil-drop dyschromia, no pitting, no crumbling) to 3 (>30 onycholysis together with oil-drop dyschromia, >50 pitting, >50% crumbling). Four features (leukonychia, splinter, hemorrhages, hyperkeratosis, and red spots in the lunula) are graded with the score of 1 = present or 0 = absent for each fingernail. Each finger has a score between 0 and 13. The total mNAPSI score is the sum of all abnormalities individual score across all fingers, and the total mNAPSI score ranges from 0 to 130. Lower numbers indicate fewer nail abnormalities. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with psoriatic nail involvement at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 25 | 25 | 30
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 25 | 25 | 29
  Change from Baseline at Week 4 | -6 (7.4) | -4 (8.5) | 0 (9.7)
  Change from Baseline at Week 8: number analyzed (Participants) | 23 | 25 | 28
  Change from Baseline at Week 8 | -7 (9.9) | -5 (11.1) | 0 (11.2)
  Change from Baseline at Week 12: number analyzed (Participants) | 24 | 25 | 28
  Change from Baseline at Week 12 | -7 (8.3) | -4 (11.7) | 1 (14.0)
  Change from Baseline at Week 16: number analyzed (Participants) | 24 | 25 | 27
  Change from Baseline at Week 16 | -8 (9.3) | -6 (9.4) | -2 (8.3)

13. Secondary Outcome: Change From Baseline in mNAPSI at Weeks 20, 24, 28, 36, and 48 in Participants With Psoriatic Nail Involvement at Baseline
Description: as for outcome 12
Time Frame: Baseline, 20, 24, 28, 36, and 48 weeks
Population: Participants in the FAS with psoriatic nail involvement at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 8 | 5
score on a scale
  Change from Baseline at Week 20: number analyzed (Participants) | 12 | 15 | 8 | 5
  Change from Baseline at Week 20 | -11 (12.3) | -5 (10.1) | -1 (4.8) | -3 (5.5)
  Change from Baseline at Week 24: number analyzed (Participants) | 12 | 13 | 6 | 5
  Change from Baseline at Week 24 | -10 (11.9) | -4 (7.5) | -2 (4.0) | -1 (1.4)
  Change from Baseline at Week 28: number analyzed (Participants) | 7 | 8 | 3 | 3
  Change from Baseline at Week 28 | -13 (15.4) | -5 (11.4) | -3 (4.9) | -3 (2.3)
  Change from Baseline at Week 36: number analyzed (Participants) | 8 | 7 | 3 | 3
  Change from Baseline at Week 36 | -13 (15.3) | -6 (8.4) | 2 (2.1) | -2 (1.2)
  Change from Baseline at Week 48: number analyzed (Participants) | 7 | 6 | 3 | 2
  Change from Baseline at Week 48 | -9 (16.6) | -3 (5.0) | 1 (5.6) | -8 (10.6)

14. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI) at Weeks 4, 8, 12, and 16 in Participants With Enthesitis at Baseline
Description: Enthesitis is assessed using LEI. The enthesitis examination by LEI evaluates the presence or absence of pain by applying local pressure on 6 anatomical sites: medial femoral condyle (left and right), lateral epicondyle (left and right), and the achilles tendon insertion (left and right). Enthesitis at each site is scored as 0 (enthesitis absent) and 1 (enthesitis present). LEI is derived as the sum of the enthesitis score over the 6 sites mentioned above. The total score ranges from 0 to 6, higher scores indicates greater degree of enthesitis. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with enthesitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 22 | 22 | 24
score on a scale
  Change from Baseline at Week 4 | 0 (1.3) | -1 (1.2) | 0 (1.9)
  Change from Baseline at Week 8: number analyzed (Participants) | 20 | 22 | 24
  Change from Baseline at Week 8 | -1 (2.4) | 0 (1.4) | 0 (1.6)
  Change from Baseline at Week 12: number analyzed (Participants) | 20 | 22 | 24
  Change from Baseline at Week 12 | -1 (2.1) | 0 (1.6) | 0 (1.5)
  Change from Baseline at Week 16: number analyzed (Participants) | 19 | 21 | 24
  Change from Baseline at Week 16 | -1 (2.4) | -1 (1.3) | 0 (1.4)
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.24, MMRM — P-value was provided from mixed-effects model for repeated measures (MMRM) having treatment, visit (categorical), treatment by visit, stratification factors, baseline value as fixed effects, participants being the random effect; LS Mean Treatment Difference = -0, 95% CI 2-sided [-1 to 0], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.22, MMRM — P-value was provided from MMRM having treatment, visit (categorical), treatment by visit, stratification factors, baseline value as fixed effects, participants being the random effect; LS Mean Treatment Difference = -1, 95% CI 2-sided [-1 to 0], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.43, MMRM — [p-value comment as in outcome 14, analysis 2]; LS Mean Treatment Difference = -0, 95% CI 2-sided [-1 to 1], Standard Error of Mean 0.5
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.70, MMRM — [p-value comment as in outcome 14, analysis 2]; LS Mean Treatment Difference = 0, 95% CI 2-sided [-1 to 1], Standard Error of Mean 0.5
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.10, MMRM — [p-value comment as in outcome 14, analysis 2]; LS Mean Treatment Difference = -1, 95% CI 2-sided [-2 to 0], Standard Error of Mean 0.5
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.90, MMRM — [p-value comment as in outcome 14, analysis 2]; LS Mean Treatment Difference = -0, 95% CI 2-sided [-1 to 1], Standard Error of Mean 0.5
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.88, MMRM — [p-value comment as in outcome 14, analysis 2]; LS Mean Treatment Difference = 0, 95% CI 2-sided [-1 to 1], Standard Error of Mean 0.5
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.89, MMRM — [p-value comment as in outcome 14, analysis 2]; LS Mean Treatment Difference = -0, 95% CI 2-sided [-1 to 1], Standard Error of Mean 0.5

15. Secondary Outcome: Change From Baseline in LEI at Weeks 20, 24, 28, 36, and 48 in Participants With Enthesitis at Baseline
Description: as for outcome 14
Time Frame: Baseline, 20, 24, 28, 36, and 48 weeks
Population: Participants in the FAS with enthesitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 9 | 5
score on a scale
  Change from Baseline at Week 20: number analyzed (Participants) | 10 | 13 | 9 | 5
  Change from Baseline at Week 20 | -2 (2.2) | -1 (1.6) | 0 (1.3) | 0 (1.8)
  Change from Baseline at Week 24: number analyzed (Participants) | 11 | 11 | 7 | 5
  Change from Baseline at Week 24 | -1 (2.0) | 0 (1.4) | 0 (0.8) | 0 (0.4)
  Change from Baseline at Week 28: number analyzed (Participants) | 6 | 7 | 4 | 4
  Change from Baseline at Week 28 | -2 (1.9) | -1 (2.2) | -1 (1.0) | 0 (0.5)
  Change from Baseline at Week 36: number analyzed (Participants) | 7 | 7 | 4 | 4
  Change from Baseline at Week 36 | -2 (1.8) | -2 (2.4) | 0 (2.1) | 0 (1.0)
  Change from Baseline at Week 48: number analyzed (Participants) | 6 | 6 | 4 | 4
  Change from Baseline at Week 48 | -3 (1.4) | -2 (2.4) | -1 (1.0) | 1 (1.3)

16. Secondary Outcome: Change From Baseline in 12-Item Psoriatic Arthritis Impact of Disease (PsAID-12) Score at Weeks 4 and 16
Description: The PsAID questionnaire assesses the impact of PsA on people's lives. The PsAID is calculated based on 12 numerical rating scales (NRS) questions. The 12 NRS is focused on pain, fatigue, skin, work and/or leisure activities, function, discomfort, sleep, coping, anxiety, embarrassment, social life, and depression. Each NRS is assessed as a number between 0 and 10. Total score is calculated as the sum of the individual scores, (some of which were multiplied by a weighting factor) divided by 20 for a total possible score of 0 to 10, where higher score indicates worse impact of disease. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | -0.97 (1.876) | -0.66 (1.492) | -0.49 (1.139)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 34
  Change from Baseline at Week 16 | -1.58 (2.263) | -1.04 (1.802) | -0.38 (1.543)

17. Secondary Outcome: Change From Baseline in PsAID-12 Score at Week 48
Description: as for outcome 16
Time Frame: Baseline, Week 48
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 17 | 19 | 10 | 8
score on a scale | -1.04 (2.441) | -1.44 (2.396) | -1.59 (1.807) | 0.39 (1.123)

18. Secondary Outcome: Percentage of Participants With PASDAS Low Disease Activity (LDA) at Weeks 4 and 16
Description: PASDAS is a composite disease activity measure for psoriatic arthritis. The PASDAS includes the following components: PGADA [using a VAS on a scale of 0 (very well) to 100 (very poor)]; PhGADA [using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity)]; 36-item short form survey (SF-36) [a questionnaire which measures quality of life across eight domains used to determine a PCS with a score range of 0-100, higher scores indicates better health status]; TJC68; SJC66; LEI [assessed at 6 sites with a score range of 0 to 6, higher scores indicates higher degree of enthesitis]; TDC [with a score range of 0 to 60, higher score indicates higher degree of dactylitis]; CRP. The score of PASDAS ranges from 0-10, lower score indicates better function. PASDAS LDA is defined as PASDAS ≤ 3.2.
Time Frame: Weeks 4 and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 4: number analyzed (Participants) | 34 | 33 | 35
  Week 4 | 8.8 [0.0 to 19.8] | 21.2 [5.7 to 36.7] | 8.6 [0.0 to 19.3]
  Week 16: number analyzed (Participants) | 31 | 33 | 33
  Week 16 | 38.7 [20.0 to 57.5] | 30.3 [13.1 to 47.5] | 12.1 [0.0 to 24.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.3, 95% CI 2-sided [-15.9 to 16.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 12.6, 95% CI 2-sided [-7.1 to 32.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 26.6, 95% CI 2-sided [3.0 to 50.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 18.2, 95% CI 2-sided [-4.1 to 40.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

19. Secondary Outcome: Percentage of Participants With PASDAS LDA at Week 48
Description: as for outcome 18
Time Frame: Week 48
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 8 | 9 | 4 | 3
percentage of participants | 50.0 [9.1 to 90.9] | 33.3 [0.0 to 69.7] | 50.0 [0.0 to 100.0] | 0 [0.0 to 16.7]

20. Secondary Outcome: Percentage of Participants Who Achieved PASDAS Remission at Weeks 4 and 16
Description: PASDAS is a composite disease activity measure for psoriatic arthritis. The PASDAS includes the following components: PGADA [using a VAS on a scale of 0 (very well) to 100 (very poor)]; PhGADA [using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity)]; 36-item short form survey (SF-36) [a questionnaire which measures quality of life across eight domains used to determine a PCS with a score range of 0-100, higher scores indicates better health status]; TJC68; SJC66; LEI [assessed at 6 sites with a score range of 0 to 6, higher scores indicates higher degree of enthesitis]; TDC [with a score range of 0 to 60, higher score indicates higher degree of dactylitis]; CRP. The score of PASDAS ranges from 0-10, lower score indicates better function. PASDAS remission is defined as PASDAS ≤ 1.9.
Time Frame: Weeks 4 and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 4: number analyzed (Participants) | 34 | 33 | 35
  Week 4 | 2.9 [0.0 to 10.1] | 0 [0.0 to 1.5] | 0 [0.0 to 1.4]
  Week 16: number analyzed (Participants) | 31 | 33 | 33
  Week 16 | 12.9 [0.0 to 26.3] | 9.1 [0.0 to 20.4] | 0 [0.0 to 1.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 2.9, 95% CI 2-sided [-5.6 to 11.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-2.9 to 2.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 12.9, 95% CI 2-sided [-2.0 to 27.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 9.1, 95% CI 2-sided [-3.7 to 21.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

21. Secondary Outcome: Percentage of Participants Who Achieved PASDAS Remission at Week 48
Description: as for outcome 20
Time Frame: Week 48
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 8 | 9 | 4 | 3
percentage of participants | 25.0 [0.0 to 61.3] | 11.1 [0.0 to 37.2] | 25.0 [0.0 to 79.9] | 0 [0.0 to 16.7]

22. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 20% Improvement Response at Weeks 2, 4, 8, 12, and 16
Description: ACR20 response is achieved when the participant has: ≥ 20% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGADA using a VAS on a scale of 0 (very well) to 100 (very poor); PHGADA using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity); HAQ-DI inclusive of activities scored on a scale of 0 (no disability) to 3 (completely disabled); HAQ-DI pain assessment using VAS on a scale of 0 (no pain) to 100 (serious pain); and hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 2: number analyzed (Participants) | 34 | 33 | 36
  Week 2 | 26.5 [10.2 to 42.8] | 6.1 [0.0 to 15.7] | 11.1 [0.0 to 22.8]
  Week 4: number analyzed (Participants) | 35 | 34 | 34
  Week 4 | 31.4 [14.6 to 48.2] | 29.4 [12.6 to 46.2] | 20.6 [5.5 to 35.7]
  Week 8: number analyzed (Participants) | 32 | 34 | 33
  Week 8 | 59.4 [40.8 to 78.0] | 32.4 [15.2 to 49.5] | 39.4 [21.2 to 57.6]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 60.6 [42.4 to 78.8] | 35.3 [17.8 to 52.8] | 32.4 [15.2 to 49.5]
  Week 16: number analyzed (Participants) | 32 | 33 | 33
  Week 16 | 56.3 [37.5 to 75.0] | 36.4 [18.4 to 54.3] | 30.3 [13.1 to 47.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.098, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 15.4, 95% CI 2-sided [-5.5 to 36.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.40, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -5.1, 95% CI 2-sided [-21.1 to 11.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.26, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 10.8, 95% CI 2-sided [-12.6 to 34.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.39, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 8.8, 95% CI 2-sided [-14.6 to 32.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.088, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 20.0, 95% CI 2-sided [-6.9 to 46.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.49, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -7.0, 95% CI 2-sided [-32.9 to 18.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.019, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 28.3, 95% CI 2-sided [2.4 to 54.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.85, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 2.9, 95% CI 2-sided [-22.5 to 28.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.036, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 25.9, 95% CI 2-sided [-0.4 to 52.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.60, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 6.1, 95% CI 2-sided [-19.7 to 31.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

23. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 20% Improvement Response at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 22
Time Frame: Weeks 18, 20, 24, 28, 36, 48, and 60
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Filgotinib 200 mg From Filgotinib 200 mg (LTE): Filgotinib 200 mg tablet orally once daily+ PTM filgotinib 100 mg tablet orally once daily for up to 44.3 weeks. Participants received filgotinib 200 mg in the Main Study.
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 15 | 18 | 7 | 7
  Week 18 | 66.7 [39.5 to 93.9] | 50.0 [24.1 to 75.9] | 42.9 [0.0 to 86.7] | 0 [0.0 to 7.1]
  Week 20: number analyzed (Participants) | 13 | 19 | 8 | 8
  Week 20 | 46.2 [15.2 to 77.1] | 47.4 [22.3 to 72.5] | 50.0 [9.1 to 90.9] | 12.5 [0.0 to 41.7]
  Week 24: number analyzed (Participants) | 13 | 16 | 4 | 6
  Week 24 | 46.2 [15.2 to 77.1] | 75.0 [50.7 to 99.3] | 0 [0.0 to 12.5] | 16.7 [0.0 to 54.8]
  Week 28: number analyzed (Participants) | 8 | 11 | 3 | 5
  Week 28 | 62.5 [22.7 to 100.0] | 72.7 [41.9 to 100.0] | 33.3 [0.0 to 100.0] | 20.0 [0.0 to 65.1]
  Week 36: number analyzed (Participants) | 9 | 10 | 3 | 4
  Week 36 | 77.8 [45.1 to 100.0] | 50.0 [14.0 to 86.0] | 0 [0.0 to 16.7] | 50.0 [0.0 to 100.0]
  Week 48: number analyzed (Participants) | 8 | 9 | 3 | 3
  Week 48 | 62.5 [22.7 to 100.0] | 44.4 [6.4 to 82.5] | 66.7 [0.0 to 100.0] | 0 [0.0 to 16.7]
  Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Week 60 | 100.0 [50.0 to 100.0] | 100.0 [50.0 to 100.0] | 100.0 [75.0 to 100.0] | 50.0 [0.0 to 100.0]

24. Secondary Outcome: Percentage of Participants Who Achieve an American College of Rheumatology 50% Improvement Response at Weeks 2, 4, 8, 12, and 16
Description: ACR50 response is achieved when the participant has: ≥ 50% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGADA using a VAS on a scale of 0 (very well) to 100 (very poor); PHGADA using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity); HAQ-DI inclusive of activities scored on a scale of 0 (no disability) to 3 (completely disabled); HAQ-DI pain assessment using VAS on a scale of 0 (no pain) to 100 (serious pain); and hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 2: number analyzed (Participants) | 34 | 33 | 36
  Week 2 | 8.8 [0.0 to 19.8] | 0 [0.0 to 1.5] | 2.8 [0.0 to 9.5]
  Week 4: number analyzed (Participants) | 36 | 34 | 35
  Week 4 | 11.1 [0.0 to 22.8] | 0 [0.0 to 1.5] | 8.6 [0.0 to 19.3]
  Week 8: number analyzed (Participants) | 32 | 34 | 33
  Week 8 | 15.6 [1.5 to 29.8] | 8.8 [0.0 to 19.8] | 9.1 [0.0 to 20.4]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 36.4 [18.4 to 54.3] | 8.8 [0.0 to 19.8] | 17.6 [3.4 to 31.9]
  Week 16: number analyzed (Participants) | 32 | 33 | 33
  Week 16 | 43.8 [25.0 to 62.5] | 18.2 [3.5 to 32.9] | 3.0 [0.0 to 10.4]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.31, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 6.0, 95% CI 2-sided [-7.8 to 19.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.48, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -2.8, 95% CI 2-sided [-11.1 to 5.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.70, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 2.5, 95% CI 2-sided [-14.1 to 19.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.17, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -8.6, 95% CI 2-sided [-20.7 to 3.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.34, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 6.5, 95% CI 2-sided [-12.5 to 25.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.98, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -0.3, 95% CI 2-sided [-16.9 to 16.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.071, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 18.7, 95% CI 2-sided [-5.1 to 42.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.27, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -8.8, 95% CI 2-sided [-27.7 to 10.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 40.7, 95% CI 2-sided [19.5 to 62.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.082, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 15.2, 95% CI 2-sided [-2.3 to 32.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

25. Secondary Outcome: Percentage of Participants Who Achieve an American College of Rheumatology 50% Improvement Response at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 24
Time Frame: Weeks 18, 20, 24, 28, 36, 48, and 60
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Filgotinib 200 mg From Placebo (LTE): Filgotinib 200 mg tablet orally once daily+ PTM filgotinib 100 mg tablet orally once daily for up to 44.1 weeks. Participants received placebo in the Main Study.
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 15 | 18 | 7 | 8
  Week 18 | 40.0 [11.9 to 68.1] | 22.2 [0.2 to 44.2] | 28.6 [0.0 to 69.2] | 0 [0.0 to 6.3]
  Week 20: number analyzed (Participants) | 13 | 19 | 8 | 8
  Week 20 | 30.8 [1.8 to 59.7] | 21.1 [0.1 to 42.0] | 25.0 [0.0 to 61.3] | 0 [0.0 to 6.3]
  Week 24: number analyzed (Participants) | 13 | 16 | 6 | 6
  Week 24 | 38.5 [8.2 to 68.8] | 56.3 [28.8 to 83.7] | 0 [0.0 to 8.3] | 0 [0.0 to 8.3]
  Week 28: number analyzed (Participants) | 8 | 11 | 3 | 5
  Week 28 | 37.5 [0.0 to 77.3] | 18.2 [0.0 to 45.5] | 0 [0.0 to 16.7] | 0 [0.0 to 10.0]
  Week 36: number analyzed (Participants) | 9 | 10 | 3 | 5
  Week 36 | 66.7 [30.3 to 100.0] | 40.0 [4.6 to 75.4] | 0 [0.0 to 16.7] | 0 [0.0 to 10.0]
  Week 48: number analyzed (Participants) | 8 | 9 | 3 | 3
  Week 48 | 50.0 [9.1 to 90.9] | 11.1 [0.0 to 37.2] | 66.7 [0.0 to 100.0] | 0 [0.0 to 16.7]
  Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Week 60 | 0 [0.0 to 50.0] | 0 [0.0 to 50.0] | 0 [0.0 to 25.0] | 50.0 [0.0 to 100.0]

26. Secondary Outcome: Percentage of Participants Who Achieve an American College of Rheumatology 70% Improvement Response at Weeks 2, 4, 8, 12, and 16
Description: ACR70 response is achieved when the participant has: ≥ 70% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGADA using a VAS on a scale of 0 (very well) to 100 (very poor); PHGADA using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity); HAQ-DI inclusive of activities scored on a scale of 0 (no disability) to 3 (completely disabled); HAQ-DI pain assessment using VAS on a scale of 0 (no pain) to 100 (serious pain); and hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with the available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 2: number analyzed (Participants) | 34 | 33 | 36
  Week 2 | 2.9 [0.0 to 10.1] | 0 [0.0 to 1.5] | 0 [0.0 to 1.4]
  Week 4: number analyzed (Participants) | 36 | 34 | 35
  Week 4 | 2.8 [0.0 to 9.5] | 0 [0.0 to 1.5] | 0 [0.0 to 1.4]
  Week 8: number analyzed (Participants) | 32 | 34 | 34
  Week 8 | 15.6 [1.5 to 29.8] | 0 [0.0 to 1.5] | 2.9 [0.0 to 10.1]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 21.2 [5.7 to 36.7] | 5.9 [0.0 to 15.3] | 2.9 [0.0 to 10.1]
  Week 16: number analyzed (Participants) | 32 | 33 | 33
  Week 16 | 12.5 [0.0 to 25.5] | 9.1 [0.0 to 20.4] | 0 [0.0 to 1.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 2.9, 95% CI 2-sided [-5.6 to 11.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-2.9 to 2.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 2.8, 95% CI 2-sided [-5.4 to 11.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-2.9 to 2.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 12.7, 95% CI 2-sided [-4.2 to 29.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -2.9, 95% CI 2-sided [-11.6 to 5.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 18.3, 95% CI 2-sided [0.2 to 36.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 2.9, 95% CI 2-sided [-9.7 to 15.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 12.5, 95% CI 2-sided [-2.0 to 27.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 9.1, 95% CI 2-sided [-3.7 to 21.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

27. Secondary Outcome: Percentage of Participants Who Achieve an American College of Rheumatology 70% Improvement Response at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 26
Time Frame: Weeks 18, 20, 24, 28, 36, 48, and 60
Population: Participants in the FAS with the available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Week 18 | 40.0 [11.9 to 68.1] | 11.1 [0.0 to 28.4] | 0 [0.0 to 6.3] | 0 [0.0 to 6.3]
  Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Week 20 | 30.8 [1.8 to 59.7] | 10.5 [0.0 to 27.0] | 0 [0.0 to 5.0] | 0 [0.0 to 6.3]
  Week 24: number analyzed (Participants) | 13 | 16 | 6 | 6
  Week 24 | 30.8 [1.8 to 59.7] | 25.0 [0.7 to 49.3] | 0 [0.0 to 8.3] | 0 [0.0 to 8.3]
  Week 28: number analyzed (Participants) | 8 | 11 | 3 | 5
  Week 28 | 37.5 [0.0 to 77.3] | 9.1 [0.0 to 30.6] | 0 [0.0 to 16.7] | 0 [0.0 to 10.0]
  Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Week 36 | 33.3 [0.0 to 69.7] | 10.0 [0.0 to 33.6] | 0 [0.0 to 12.5] | 0 [0.0 to 10.0]
  Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Week 48 | 25.0 [0.0 to 61.3] | 11.1 [0.0 to 37.2] | 0 [0.0 to 12.5] | 0 [0.0 to 16.7]
  Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Week 60 | 0 [0.0 to 50.0] | 0 [0.0 to 50.0] | 0 [0.0 to 25.0] | 0 [0.0 to 25.0]

28. Secondary Outcome: Change From Baseline in Individual ACR Component: Tender Joint Count Based on 68 Joints (TJC68) at Weeks 2, 4, 8, 12, and 16
Description: TJC68 is an assessment of 68 joints. Each joint is evaluated as 'normal', 'tender', 'tender and swollen', or 'not able to evaluate'. It is derived as the sum of all tender joints. The overall tender joint count ranged from 0 to 68, with a higher score indicating a greater degree of tenderness. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
tender joint count
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 33 | 36
  Change from Baseline at Week 2 | -6 (10.3) | -5 (12.2) | -2 (11.9)
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | -7 (10.7) | -7 (10.2) | -4 (13.9)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 34
  Change from Baseline at Week 8 | -10 (13.2) | -8 (11.5) | -8 (13.2)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 34
  Change from Baseline at Week 12 | -12 (15.4) | -10 (12.7) | -9 (10.7)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 33
  Change from Baseline at Week 16 | -13 (15.7) | -11 (12.5) | -10 (10.7)

29. Secondary Outcome: Change From Baseline in Individual ACR Component: TJC68 at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 28
Time Frame: Baseline, 18, 20, 24, 28, 36, 48, and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
tender joint count
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -12 (14.8) | -12 (9.9) | -4 (4.6) | -2 (6.4)
  Change from Baseline at Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Change from Baseline at Week 20 | -18 (18.7) | -10 (12.2) | -4 (5.7) | 1 (8.9)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Change from Baseline at Week 24 | -16 (25.6) | -11 (12.0) | -1 (2.3) | -1 (12.1)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Change from Baseline at Week 28 | -21 (20.0) | -14 (14.2) | 0 (1.3) | -2 (13.4)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -25 (19.6) | -13 (12.3) | 0 (1.9) | -5 (10.8)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -22 (21.6) | -17 (14.7) | -6 (9.9) | -3 (14.0)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | -60 (NA) — SD cannot be calculated for 1 participant | -11 (NA) — SD cannot be calculated for 1 participant | -5 (3.5) | 3 (17.7)

30. Secondary Outcome: Change From Baseline in ACR Component: Swollen Joint Count Based on 66 Joints (SJC66) at Weeks 2, 4, 8, 12, and 16
Description: SJC66 is an assessment of 66 joints. Each joint was evaluated as 'normal', 'swollen', 'tender and swollen', or 'not able to evaluate'. It is derived as the sum of all swollen joints. The overall swollen joint count ranged from 0 to 66, with a higher score indicating a greater degree of swelling. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
swollen joint count
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 33 | 36
  Change from Baseline at Week 2 | -3 (7.4) | -3 (5.6) | 0 (6.5)
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | -6 (7.1) | -3 (4.4) | -3 (6.0)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 34
  Change from Baseline at Week 8 | -7 (8.5) | -4 (5.0) | -4 (6.3)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 34
  Change from Baseline at Week 12 | -8 (8.6) | -4 (7.2) | -4 (5.9)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 33
  Change from Baseline at Week 16 | -7 (7.6) | -6 (6.9) | -5 (6.1)

31. Secondary Outcome: Change From Baseline in ACR Component: SJC66 at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 30
Time Frame: Baseline, 18, 20, 24, 28, 36, 48, and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joint count
Groups:
- Filgotinib 100 mg From Placebo (LTE): Filgotinib 100 mg tablet orally once daily+ PTM filgotinib 200 mg tablet orally once daily for up to 44 weeks. Participants received placebo in the Main Study.
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
swollen joint count
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -10 (7.7) | -8 (7.6) | -3 (3.2) | -1 (2.6)
  Change from Baseline at Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Change from Baseline at Week 20 | -11 (9.5) | -6 (6.0) | -3 (4.2) | 2 (6.6)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Change from Baseline at Week 24 | -10 (9.9) | -6 (4.0) | -2 (4.1) | -1 (2.1)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Change from Baseline at Week 28 | -14 (7.8) | -6 (4.2) | 0 (0.5) | 2 (6.9)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -14 (7.1) | -7 (4.3) | -2 (3.3) | -1 (3.4)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -13 (9.5) | -7 (4.1) | -6 (8.9) | 2 (4.9)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | -21 (NA) — SD cannot be calculated for 1 participant. | -2 (NA) — SD cannot be calculated for 1 participant. | -5 (2.8) | 2 (7.1)

32. Secondary Outcome: Change From Baseline in Individual ACR Component: Patient's Global Assessment of Disease Activity (PGADA) at Weeks 2, 4, 8, 12, and 16
Description: PGADA is assessed by the participants using a VAS on a scale of 0 (very well) to 100 (very poor). A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 33 | 36
  Change from Baseline at Week 2 | -13 (24.3) | -7 (18.6) | -4 (21.6)
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | -9 (27.2) | -8 (19.2) | -9 (20.6)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 34
  Change from Baseline at Week 8 | -20 (28.6) | -7 (21.9) | -11 (23.0)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 34
  Change from Baseline at Week 12 | -24 (32.4) | -11 (19.4) | -8 (23.2)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 33
  Change from Baseline at Week 16 | -21 (30.3) | -13 (24.2) | -5 (25.7)

33. Secondary Outcome: Change From Baseline in Individual ACR Component: PGADA at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 32
Time Frame: Baseline, 18, 20, 24, 28, 36, 48, and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
score on a scale
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -24 (26.8) | -20 (25.4) | -13 (16.4) | -11 (21.5)
  Change from Baseline at Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Change from Baseline at Week 20 | -16 (30.0) | -18 (31.0) | -15 (25.3) | -9 (25.1)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Change from Baseline at Week 24 | -12 (30.2) | -28 (34.3) | -19 (26.4) | -18 (9.8)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Change from Baseline at Week 28 | -19 (27.9) | -24 (30.4) | -10 (34.0) | -21 (9.5)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -26 (27.5) | -21 (30.6) | 11 (34.9) | -24 (8.6)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -31 (17.0) | -23 (27.6) | -18 (21.6) | -6 (5.1)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | -32 (NA) — SD cannot be calculated for 1 participant. | -10 (NA) — SD cannot be calculated for 1 participant. | -14 (18.4) | -6 (12.0)

34. Secondary Outcome: Change From Baseline in Individual ACR Component: Physician's Global Assessment of Disease Activity (PhGADA) at Weeks 2, 4, 8, 12, and 16
Description: PhGADA is assessed by the physician using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 32 | 36
  Change from Baseline at Week 2 | -14 (21.1) | -16 (14.5) | -8 (16.0)
  Change from Baseline at Week 4: number analyzed (Participants) | 35 | 33 | 35
  Change from Baseline at Week 4 | -20 (21.3) | -19 (15.8) | -12 (18.5)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 34
  Change from Baseline at Week 8 | -31 (22.8) | -24 (14.1) | -17 (20.1)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 33
  Change from Baseline at Week 12 | -34 (21.2) | -25 (17.9) | -15 (19.5)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 33
  Change from Baseline at Week 16 | -35 (24.5) | -27 (20.3) | -18 (20.9)

35. Secondary Outcome: Change From Baseline in Individual ACR Component: PhGADA at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 34
Time Frame: Baseline, 18, 20, 24, 28, 36, 48, and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
score on a scale
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -36 (24.0) | -29 (17.7) | -7 (14.0) | -6 (10.7)
  Change from Baseline at Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Change from Baseline at Week 20 | -32 (28.8) | -29 (15.4) | -14 (11.9) | -7 (8.9)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Change from Baseline at Week 24 | -40 (24.8) | -29 (15.1) | -21 (15.0) | -8 (5.0)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Change from Baseline at Week 28 | -43 (16.8) | -35 (14.4) | -27 (19.1) | -3 (22.3)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -47 (19.6) | -37 (13.2) | -20 (13.1) | -8 (7.2)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -46 (23.8) | -31 (12.9) | -25 (4.0) | -1 (2.3)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | -77 (NA) — SD cannot be calculated for 1 participant | -33 (NA) — SD cannot be calculated for 1 participant | -18 (13.4) | -16 (4.2)

36. Secondary Outcome: Change From Baseline in Individual ACR Component: Health Assessment Questionnaire Disability Index (HAQ-DI)'s Pain Assessment at Weeks 2, 4, 8, 12, and 16
Description: HAQ-DI's pain assessment is done using VAS on a scale of 0 (no pain) to 100 (serious pain). A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 33 | 36
  Change from Baseline at Week 2 | -10 (20.4) | -3 (12.0) | -4 (14.7)
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | -10 (23.0) | -4 (17.0) | -8 (19.1)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 34
  Change from Baseline at Week 8 | -17 (22.7) | -8 (21.3) | -12 (20.0)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 34
  Change from Baseline at Week 12 | -24 (30.0) | -12 (22.2) | -6 (21.9)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 33
  Change from Baseline at Week 16 | -22 (26.4) | -13 (21.7) | -6 (23.5)

37. Secondary Outcome: Change From Baseline in Individual ACR Component: Health Assessment Questionnaire Disability Index (HAQ-DI)'s Pain Assessment at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 36
Time Frame: Baseline, 18, 20, 24, 28, 36, 48, and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
score on a scale
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -26 (26.3) | -13 (24.7) | -18 (25.5) | -7 (8.5)
  Change from Baseline at Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Change from Baseline at Week 20 | -13 (30.3) | -18 (24.5) | -19 (24.5) | -7 (23.5)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Change from Baseline at Week 24 | -18 (30.0) | -25 (29.4) | -17 (22.0) | -12 (12.7)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Change from Baseline at Week 28 | -23 (20.7) | -19 (26.6) | -21 (25.0) | -21 (4.2)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -27 (23.7) | -24 (23.4) | -2 (25.4) | -17 (8.4)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -30 (22.4) | -23 (28.0) | -24 (23.6) | -8 (5.5)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | -22 (NA) — SD cannot be calculated for 1 participant. | -35 (NA) — SD cannot be calculated for 1 participant. | -20 (28.3) | -23 (2.8)

38. Secondary Outcome: Change From Baseline in Individual ACR Component: High-Sensitivity C- Reactive Protein (hsCRP) at Weeks 2, 4, 8, 12, and 16
Description: The hsCRP is the ACR core set measure of acute phase reactant. It was measured at the central laboratory to help assess the effect of filgotinib on the participant's psoriatic arthritis. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
mg/L
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 33 | 35
  Change from Baseline at Week 2 | -4.01 (6.669) | 0.53 (14.972) | 0.56 (8.836)
  Change from Baseline at Week 4: number analyzed (Participants) | 35 | 34 | 34
  Change from Baseline at Week 4 | -4.42 (10.769) | -1.20 (6.309) | 0.05 (5.566)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 33
  Change from Baseline at Week 8 | -5.21 (16.030) | -1.68 (5.085) | -1.35 (11.841)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 33
  Change from Baseline at Week 12 | -4.57 (12.585) | -2.43 (6.248) | -1.09 (11.687)
  Change from Baseline at Week 16: number analyzed (Participants) | 31 | 33 | 32
  Change from Baseline at Week 16 | -4.96 (13.906) | -0.05 (7.210) | -0.37 (13.337)

39. Secondary Outcome: Change From Baseline in Individual ACR Component: hsCRP at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 38
Time Frame: Baseline, 18, 20, 24, 28, 36, 48, and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Filgotinib 200 mg From Placebo (LTE): Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet for orally once daily up to 44.1 weeks. Participants received placebo in the Main Study.
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
mg/L
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -1.49 (5.017) | -0.70 (4.064) | -3.54 (6.980) | -3.05 (2.871)
  Change from Baseline at Week 20: number analyzed (Participants) | 14 | 19 | 10 | 8
  Change from Baseline at Week 20 | -0.68 (4.040) | -1.36 (4.214) | -3.83 (6.244) | -2.49 (3.285)
  Change from Baseline at Week 24: number analyzed (Participants) | 14 | 16 | 7 | 7
  Change from Baseline at Week 24 | -3.31 (5.963) | -2.21 (4.515) | -1.01 (5.187) | -1.72 (4.828)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 4
  Change from Baseline at Week 28 | 1.56 (6.011) | -0.92 (5.460) | 2.24 (7.159) | -2.33 (2.777)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -3.10 (5.507) | -0.84 (7.796) | -1.92 (1.217) | -2.38 (1.959)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -1.84 (6.262) | 0.07 (6.378) | -2.08 (2.353) | -1.68 (1.992)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | -1.65 (NA) — SD cannot be calculated for 1 participant. | -12.32 (NA) — SD cannot be calculated for 1 participant. | 2.39 (4.851) | -2.73 (0.827)

40. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) C-Reactive Protein (CRP) at Weeks 2, 4, 8, 12, and 16
Description: The DAS28(CRP) is a measure of the participant's disease activity calculated using the tender joint count (28 joints), swollen joint count (28 joints), PGADA [using a VAS on a scale of 0 (very well) to 100 (very poor)] and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 33 | 35
  Change from Baseline at Week 2 | -1.0 (1.09) | -0.7 (0.69) | -0.2 (0.70)
  Change from Baseline at Week 4: number analyzed (Participants) | 35 | 34 | 34
  Change from Baseline at Week 4 | -1.2 (1.18) | -0.7 (0.78) | -0.7 (1.18)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 33
  Change from Baseline at Week 8 | -1.5 (1.18) | -1.1 (0.99) | -1.1 (1.41)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 33
  Change from Baseline at Week 12 | -1.8 (1.37) | -1.3 (1.21) | -1.0 (1.10)
  Change from Baseline at Week 16: number analyzed (Participants) | 31 | 33 | 32
  Change from Baseline at Week 16 | -1.7 (1.35) | -1.3 (1.04) | -1.0 (1.26)

41. Secondary Outcome: Change From Baseline in DAS28(CRP) at Weeks 18, 20, 24, 28, 36, 48 and 60
Description: as for outcome 40
Time Frame: Baseline, 18, 20, 24, 28, 36, 48 and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
score on a scale
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -2.1 (1.37) | -1.8 (0.84) | -0.9 (0.70) | -0.4 (0.92)
  Change from Baseline at Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Change from Baseline at Week 20 | -1.9 (1.34) | -1.7 (0.90) | -1.1 (0.71) | -0.2 (1.34)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Change from Baseline at Week 24 | -1.8 (1.75) | -1.9 (1.13) | -0.8 (0.66) | -0.7 (1.37)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 4
  Change from Baseline at Week 28 | -2.1 (1.10) | -2.2 (0.84) | -0.9 (0.73) | -0.5 (1.79)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -2.9 (1.38) | -2.1 (1.00) | -0.6 (1.30) | -0.5 (1.10)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -2.7 (1.37) | -2.2 (0.93) | -1.3 (0.67) | 0.5 (1.62)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | -4.9 (NA) — SD cannot be calculated for 1 participant. | -0.4 (NA) — SD cannot be calculated for 1 participant. | -0.7 (0.14) | 0.1 (2.61)

42. Secondary Outcome: Percentage of Participants Who Achieved DAS28(CRP) LDA at Weeks 2, 4, 8, 12, and 16
Description: The DAS28 (CRP) is a measure of the participant's disease activity calculated using the tender joint count (28 joints), swollen joint count (28 joints), PGADA (VAS; 0 = very well to 100 = very poor), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. DAS28 (CRP) LDA is defined as DAS28(CRP) ≤ 3.2.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 2: number analyzed (Participants) | 34 | 33 | 36
  Week 2 | 20.6 [5.5 to 35.7] | 18.2 [3.5 to 32.9] | 11.1 [0.0 to 22.8]
  Week 4: number analyzed (Participants) | 35 | 34 | 35
  Week 4 | 40.0 [22.3 to 57.7] | 26.5 [10.2 to 42.8] | 20.0 [5.3 to 34.7]
  Week 8: number analyzed (Participants) | 32 | 34 | 34
  Week 8 | 53.1 [34.3 to 72.0] | 38.2 [20.4 to 56.0] | 35.3 [17.8 to 52.8]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 51.5 [32.9 to 70.1] | 41.2 [23.2 to 59.2] | 26.5 [10.2 to 42.8]
  Week 16: number analyzed (Participants) | 31 | 33 | 33
  Week 16 | 54.8 [35.7 to 74.0] | 42.4 [24.0 to 60.8] | 36.4 [18.4 to 54.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 9.5, 95% CI 2-sided [-10.4 to 29.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 7.1, 95% CI 2-sided [-12.5 to 26.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 20.0, 95% CI 2-sided [-3.8 to 43.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 6.5, 95% CI 2-sided [-16.3 to 29.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 17.8, 95% CI 2-sided [-8.8 to 44.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 2.9, 95% CI 2-sided [-22.9 to 28.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 25.0, 95% CI 2-sided [-0.5 to 50.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 14.7, 95% CI 2-sided [-10.5 to 39.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 18.5, 95% CI 2-sided [-8.7 to 45.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 6.1, 95% CI 2-sided [-20.5 to 32.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

43. Secondary Outcome: Percentage of Participants Who Achieved DAS28(CRP) LDA at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 42
Time Frame: Weeks 18, 20, 24, 28, 36, 48, and 60
Population: Participants in FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Week 18 | 60.0 [31.9 to 88.1] | 66.7 [42.1 to 91.2] | 62.5 [22.7 to 100.0] | 50.0 [9.1 to 90.9]
  Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Week 20 | 38.5 [8.2 to 68.8] | 47.4 [22.3 to 72.5] | 100.0 [95.0 to 100.0] | 37.5 [0.0 to 77.3]
  Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Week 24 | 38.5 [8.2 to 68.8] | 75.0 [50.7 to 99.3] | 71.4 [30.8 to 100.0] | 71.4 [30.8 to 100.0]
  Week 28: number analyzed (Participants) | 8 | 11 | 4 | 4
  Week 28 | 50.0 [9.1 to 90.9] | 100.0 [95.5 to 100.0] | 100.0 [87.5 to 100.0] | 25.0 [0.0 to 79.9]
  Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Week 36 | 77.8 [45.1 to 100.0] | 90.0 [66.4 to 100.0] | 50.0 [0.0 to 100.0] | 40.0 [0.0 to 92.9]
  Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Week 48 | 75.0 [38.7 to 100.0] | 88.9 [62.8 to 100.0] | 100.0 [87.5 to 100.0] | 0 [0.0 to 16.7]
  Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Week 60 | 100.0 [50.0 to 100.0] | 0 [0.0 to 50.0] | 50.0 [0.0 to 100.0] | 50.0 [0.0 to 100.0]

44. Secondary Outcome: Percentage of Participants Who Achieved DAS28(CRP) Remission at Weeks 2, 4, 8, 12, and 16
Description: The DAS28 (CRP) is a measure of the participant's disease activity calculated using the tender joint count (28 joints), swollen joint count (28 joints), PGADA (VAS; 0 = very well to 100 = very poor), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. DAS28 (CRP) remission is defined as DAS28 (CRP) < 2.6.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in FAS with the available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 2: number analyzed (Participants) | 34 | 33 | 36
  Week 2 | 11.8 [0.0 to 24.1] | 6.1 [0.0 to 15.7] | 2.8 [0.0 to 9.5]
  Week 4: number analyzed (Participants) | 35 | 34 | 35
  Week 4 | 20.0 [5.3 to 34.7] | 8.8 [0.0 to 19.8] | 14.3 [1.3 to 27.3]
  Week 8: number analyzed (Participants) | 32 | 34 | 34
  Week 8 | 21.9 [6.0 to 37.8] | 20.6 [5.5 to 35.7] | 20.6 [5.5 to 35.7]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 33.3 [15.7 to 50.9] | 32.4 [15.2 to 49.5] | 11.8 [0.0 to 24.1]
  Week 16: number analyzed (Participants) | 31 | 33 | 33
  Week 16 | 38.7 [20.0 to 57.5] | 24.2 [8.1 to 40.4] | 21.2 [5.7 to 36.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 9.0, 95% CI 2-sided [-6.0 to 23.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 3.3, 95% CI 2-sided [-9.4 to 15.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 5.7, 95% CI 2-sided [-14.7 to 26.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = -5.5, 95% CI 2-sided [-23.4 to 12.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 1.3, 95% CI 2-sided [-21.5 to 24.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-22.2 to 22.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 21.6, 95% CI 2-sided [-0.8 to 43.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 20.6, 95% CI 2-sided [-1.4 to 42.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 17.5, 95% CI 2-sided [-7.7 to 42.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 3.0, 95% CI 2-sided [-20.2 to 26.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

45. Secondary Outcome: Percentage of Participants Who Achieved DAS28(CRP) Remission at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 44
Time Frame: Weeks 18, 20, 24, 28, 36, 48, and 60
Population: Participants in FAS with the available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Week 18 | 53.3 [24.8 to 81.9] | 44.4 [18.7 to 70.2] | 62.5 [22.7 to 100.0] | 25.0 [0.0 to 61.3]
  Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Week 20 | 30.8 [1.8 to 59.7] | 31.6 [8.0 to 55.1] | 60.0 [24.6 to 95.4] | 25.0 [0.0 to 61.3]
  Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Week 24 | 38.5 [8.2 to 68.8] | 62.5 [35.7 to 89.3] | 57.1 [13.3 to 100.0] | 42.9 [0.0 to 86.7]
  Week 28: number analyzed (Participants) | 8 | 11 | 4 | 4
  Week 28 | 50.0 [9.1 to 90.9] | 63.6 [30.7 to 96.6] | 75.0 [20.1 to 100.0] | 25.0 [0.0 to 79.9]
  Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Week 36 | 55.6 [17.5 to 93.6] | 50.0 [14.0 to 86.0] | 50.0 [0.0 to 100.0] | 20.0 [0.0 to 65.1]
  Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Week 48 | 62.5 [22.7 to 100.0] | 55.6 [17.5 to 93.6] | 100.0 [87.5 to 100.0] | 0 [0.0 to 16.7]
  Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Week 60 | 100.0 [50.0 to 100.0] | 0 [0.0 to 50.0] | 50.0 [0.0 to 100.0] | 50.0 [0.0 to 100.0]

46. Secondary Outcome: Time to Achieve DAS28(CRP) LDA
Description: The DAS28 (CRP) is a measure of the participant's disease activity calculated using the TJC (28 joints), SJC (28 joints), PGADA (VAS; 0 = very well to 100 = very poor), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. DAS28 (CRP) LDA is defined as DAS28 (CRP) ≤ 3.2. Time to achieve DAS28(CRP) LDA is the number of days from the first dose date of study drug administration to the first time when a participant achieves DAS28(CRP) LDA.
Time Frame: Approximately 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 34 | 32 | 35
days | 57 [29 to 113] | NA [30 to NA] — Median and Upper Inter-Quartile Range was not estimable due to the low number of participants with DAS28(CRP) LDA. | 115 [56 to NA] — Median and Upper Inter-Quartile Range was not estimable due to the low number of participants with DAS28(CRP) LDA.

47. Secondary Outcome: Percentage of Participants Who Achieved DAPSA LDA at Weeks 2, 4, 8, 12, and 16
Description: DAPSA is calculated by summing the following components: TJC68; SJC66; PGADA [using VAS on a scale of 0 (very well) to 100 very poor)]; PGAPI [using a VAS on a scale of 0 (no pain) to 100 (serious pain)] and CRP. DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. DAPSA LDA is defined as DAPSA ≤ 14.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 2: number analyzed (Participants) | 34 | 33 | 36
  Week 2 | 17.6 [3.4 to 31.9] | 12.1 [0.0 to 24.8] | 8.3 [0.0 to 18.8]
  Week 4: number analyzed (Participants) | 35 | 34 | 35
  Week 4 | 25.7 [9.8 to 41.6] | 17.6 [3.4 to 31.9] | 20.0 [5.3 to 34.7]
  Week 8: number analyzed (Participants) | 32 | 34 | 34
  Week 8 | 40.6 [22.0 to 59.2] | 29.4 [12.6 to 46.2] | 35.3 [17.8 to 52.8]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 51.5 [32.9 to 70.1] | 41.2 [23.2 to 59.2] | 32.4 [15.2 to 49.5]
  Week 16: number analyzed (Participants) | 31 | 33 | 33
  Week 16 | 54.8 [35.7 to 74.0] | 39.4 [21.2 to 57.6] | 36.4 [18.4 to 54.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 9.3, 95% CI 2-sided [-9.2 to 27.8]
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 3.8, 95% CI 2-sided [-13.5 to 21.0]
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 5.7, 95% CI 2-sided [-16.8 to 28.2]
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = -2.4, 95% CI 2-sided [-23.7 to 19.0]
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 5.3, 95% CI 2-sided [-21.1 to 31.8]
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -5.9, 95% CI 2-sided [-31.0 to 19.3]
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 19.2, 95% CI 2-sided [-7.0 to 45.3]
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 8.8, 95% CI 2-sided [-16.9 to 34.6]
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 18.5, 95% CI 2-sided [-8.7 to 45.6]
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 3.0, 95% CI 2-sided [-23.4 to 29.5]

48. Secondary Outcome: Percentage of Participants Who Achieved DAPSA LDA at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 47
Time Frame: Weeks 18, 20, 24, 28, 36, 48, and 60
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Week 18 | 53.3 [24.8 to 81.9] | 50.0 [24.1 to 75.9] | 75.0 [38.7 to 100.0] | 50.0 [9.1 to 90.9]
  Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Week 20 | 30.8 [1.8 to 59.7] | 47.4 [22.3 to 72.5] | 80.0 [50.2 to 100.0] | 37.5 [0.0 to 77.3]
  Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Week 24 | 38.5 [8.2 to 68.8] | 75.0 [50.7 to 99.3] | 71.4 [30.8 to 100.0] | 42.9 [0.0 to 86.7]
  Week 28: number analyzed (Participants) | 8 | 11 | 4 | 4
  Week 28 | 62.5 [22.7 to 100.0] | 72.7 [41.9 to 100.0] | 100.0 [87.5 to 100.0] | 50.0 [0.0 to 100.0]
  Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Week 36 | 66.7 [30.3 to 100.0] | 60.0 [24.6 to 95.4] | 50.0 [0.0 to 100.0] | 60.0 [7.1 to 100.0]
  Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Week 48 | 62.5 [22.7 to 100.0] | 77.8 [45.1 to 100.0] | 75.0 [20.1 to 100.0] | 33.3 [0.0 to 100.0]
  Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Week 60 | 0 [0.0 to 50.0] | 0 [0.0 to 50.0] | 50.0 [0.0 to 100.0] | 50.0 [0.0 to 100.0]

49. Secondary Outcome: Percentage of Participants Who Achieved DAPSA Remission at Weeks 2, 4, 8, 12, and 16
Description: DAPSA is calculated by summing the following components: TJC68; SJC66; PGADA [using VAS on a scale of 0 (very well) to 100 very poor)]; PGAPI [using a VAS on a scale of 0 (no pain) to 100 (serious pain)] and CRP. DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. DAPSA remission is defined as DAPSA ≤ 4.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 2: number analyzed (Participants) | 34 | 33 | 36
  Week 2 | 0 [0.0 to 1.5] | 3.0 [0.0 to 10.4] | 2.8 [0.0 to 9.5]
  Week 4: number analyzed (Participants) | 35 | 34 | 35
  Week 4 | 2.9 [0.0 to 9.8] | 0 [0.0 to 1.5] | 5.7 [0.0 to 14.8]
  Week 8: number analyzed (Participants) | 32 | 34 | 34
  Week 8 | 9.4 [0.0 to 21.0] | 2.9 [0.0 to 10.1] | 8.8 [0.0 to 19.8]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 15.2 [1.4 to 28.9] | 5.9 [0.0 to 15.3] | 2.9 [0.0 to 10.1]
  Week 16: number analyzed (Participants) | 31 | 33 | 33
  Week 16 | 16.1 [1.6 to 30.7] | 15.2 [1.4 to 28.9] | 3.0 [0.0 to 10.4]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = -2.8, 95% CI 2-sided [-11.0 to 5.4]
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 0.3, 95% CI 2-sided [-10.6 to 11.1]
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = -2.9, 95% CI 2-sided [-15.2 to 9.5]
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = -5.7, 95% CI 2-sided [-16.3 to 4.9]
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 0.6, 95% CI 2-sided [-16.4 to 17.5]
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -5.9, 95% CI 2-sided [-19.9 to 8.2]
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 12.2, 95% CI 2-sided [-4.3 to 28.7]
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 2.9, 95% CI 2-sided [-9.7 to 15.6]
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 13.1, 95% CI 2-sided [-4.2 to 30.4]
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 12.1, 95% CI 2-sided [-4.5 to 28.7]

50. Secondary Outcome: Percentage of Participants Who Achieved DAPSA Remission at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 49
Time Frame: Weeks 18, 20, 24, 28, 36, 48, and 60
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Week 18 | 46.7 [18.1 to 75.2] | 16.7 [0.0 to 36.7] | 50.0 [9.1 to 90.9] | 12.5 [0.0 to 41.7]
  Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Week 20 | 23.1 [0.0 to 49.8] | 15.8 [0.0 to 34.8] | 20.0 [0.0 to 49.8] | 0 [0.0 to 6.3]
  Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Week 24 | 30.8 [1.8 to 59.7] | 43.8 [16.3 to 71.2] | 28.6 [0.0 to 69.2] | 14.3 [0.0 to 47.4]
  Week 28: number analyzed (Participants) | 8 | 11 | 4 | 4
  Week 28 | 37.5 [0.0 to 77.3] | 18.2 [0.0 to 45.5] | 50.0 [0.0 to 100.0] | 0 [0.0 to 12.5]
  Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Week 36 | 55.6 [17.5 to 93.6] | 10.0 [0.0 to 33.6] | 25.0 [0.0 to 79.9] | 0 [0.0 to 10.0]
  Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Week 48 | 50.0 [9.1 to 90.9] | 22.2 [0.0 to 54.9] | 75.0 [20.1 to 100.0] | 0 [0.0 to 16.7]
  Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Week 60 | 0 [0.0 to 50.0] | 0 [0.0 to 50.0] | 50.0 [0.0 to 100.0] | 0 [0.0 to 25.0]

51. Secondary Outcome: Time to Achieve DAPSA LDA
Description: DAPSA is calculated by summing the following components: TJC68; SJC66; PGADA [using VAS on a scale of 0 (very well) to 100 very poor)]; PGAPI [using a VAS on a scale of 0 (no pain) to 100 (serious pain)] and CRP. DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. DAPSA LDA is defined as DAPSA ≤ 14. Time to achieve DAPSA LDA is the number of days from the first dose date of study drug administration to the first time when a participant achieves DAPSA LDA. If the DAPSA LDA is not achieved during main study phase, the time to achieve DAPSA LDA will be censored at the last non-missing DAPSA LDA assessment date during main study phase. If the component scores of DAPSA LDA are at different dates for a visit, the latest date will be used for the derivation of time to achieve DAPSA LDA.
Time Frame: Approximately 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 33 | 35
days | 84 [29 to 114] | NA [58 to NA] — Median and Upper Inter-Quartile Range was not estimable due to the low number of participants with DAPSA LDA. | NA [55 to NA] — Median and Upper Inter-Quartile Range was not estimable due to the low number of participants with DAPSA LDA.

52. Secondary Outcome: Percentage of Participants Who Achieved Psoriatic Arthritis Response Criteria (PsARC) Response at Weeks 2, 4, 8, 12, and 16
Description: The PsARC response was defined as improvement in at least 2 of the following 4 criteria; ≥ 30% decrease in SJC66, ≥ 30% decrease in TJC68, ≥ 20% decrease in PGADA (VAS; 0 = very well to 100 = very poor), ≥ 20% decrease in PhGADA (VAS; 0 = no disease activity to 100 = maximum disease activity) and with at least one of the 2 joint criteria, with no deterioration in any other criteria.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
percentage of participants
  Week 2: number analyzed (Participants) | 34 | 33 | 36
  Week 2 | 32.4 [15.2 to 49.5] | 21.2 [5.7 to 36.7] | 13.9 [1.2 to 26.6]
  Week 4: number analyzed (Participants) | 36 | 34 | 35
  Week 4 | 41.7 [24.2 to 59.2] | 41.2 [23.2 to 59.2] | 25.7 [9.8 to 41.6]
  Week 8: number analyzed (Participants) | 32 | 34 | 34
  Week 8 | 68.8 [51.1 to 86.4] | 44.1 [26.0 to 62.3] | 50.0 [31.7 to 68.3]
  Week 12: number analyzed (Participants) | 33 | 34 | 34
  Week 12 | 75.8 [59.6 to 91.9] | 58.8 [40.8 to 76.8] | 35.3 [17.8 to 52.8]
  Week 16: number analyzed (Participants) | 32 | 33 | 33
  Week 16 | 62.5 [44.2 to 80.8] | 48.5 [29.9 to 67.1] | 42.4 [24.0 to 60.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 18.5, 95% CI 2-sided [-3.8 to 40.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 7.3, 95% CI 2-sided [-13.5 to 28.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 16.0, 95% CI 2-sided [-8.5 to 40.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 15.5, 95% CI 2-sided [-9.4 to 40.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 18.8, 95% CI 2-sided [-7.5 to 45.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -5.9, 95% CI 2-sided [-32.5 to 20.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 40.5, 95% CI 2-sided [15.8 to 65.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 23.5, 95% CI 2-sided [-2.5 to 49.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 20.1, 95% CI 2-sided [-6.8 to 46.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 6.1, 95% CI 2-sided [-21.0 to 33.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

53. Secondary Outcome: Percentage of Participants Who Achieved PsARC Response at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 52
Time Frame: Weeks 18, 20, 24, 28, 36, 48, and 60
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 15 | 18 | 7 | 7
  Week 18 | 73.3 [47.6 to 99.0] | 83.3 [63.3 to 100.0] | 42.9 [0.0 to 86.7] | 28.6 [0.0 to 69.2]
  Week 20: number analyzed (Participants) | 13 | 19 | 9 | 7
  Week 20 | 61.5 [31.2 to 91.8] | 68.4 [44.9 to 92.0] | 44.4 [6.4 to 82.5] | 28.6 [0.0 to 69.2]
  Week 24: number analyzed (Participants) | 13 | 16 | 6 | 6
  Week 24 | 53.8 [22.9 to 84.8] | 68.8 [42.9 to 94.6] | 16.7 [0.0 to 54.8] | 16.7 [0.0 to 54.8]
  Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Week 28 | 75.0 [38.7 to 100.0] | 63.6 [30.7 to 96.6] | 50.0 [0.0 to 100.0] | 0 [0.0 to 10.0]
  Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Week 36 | 88.9 [62.8 to 100.0] | 70.0 [36.6 to 100.0] | 25.0 [0.0 to 79.9] | 20.0 [0.0 to 65.1]
  Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Week 48 | 87.5 [58.3 to 100.0] | 66.7 [30.3 to 100.0] | 100.0 [87.5 to 100.0] | 0 [0.0 to 16.7]
  Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Week 60 | 100.0 [50.0 to 100.0] | 100.0 [50.0 to 100.0] | 50.0 [0.0 to 100.0] | 0 [0.0 to 25.0]

54. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, where 0 = none, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). A higher score indicates more severe disease. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 16 | 17 | 16
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 16 | 17 | 15
  Change from Baseline at Week 4 | -1.8 (2.79) | -2.0 (3.70) | -1.5 (7.87)
  Change from Baseline at Week 8: number analyzed (Participants) | 16 | 17 | 14
  Change from Baseline at Week 8 | -3.6 (4.82) | -1.7 (5.27) | -4.3 (6.30)
  Change from Baseline at Week 12: number analyzed (Participants) | 16 | 17 | 14
  Change from Baseline at Week 12 | -4.5 (6.79) | -2.3 (5.28) | -4.9 (7.10)
  Change from Baseline at Week 16: number analyzed (Participants) | 15 | 17 | 14
  Change from Baseline at Week 16 | -5.5 (6.90) | -1.0 (7.34) | -5.4 (6.10)

55. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) at Weeks 20, 24, 28, 36, and 48 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, where 0 = none, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). A higher score indicates more severe disease. A negative change from baseline indicates improvement.
Time Frame: Baseline, 20, 24, 28, 36, and 48 weeks
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 16 | 17 | 5 | 2
score on a scale
  Change from Baseline at Week 20: number analyzed (Participants) | 8 | 7 | 5 | 2
  Change from Baseline at Week 20 | -0.4 (7.20) | -2.9 (3.83) | -2.0 (2.21) | -1.3 (1.84)
  Change from Baseline at Week 24: number analyzed (Participants) | 7 | 7 | 4 | 2
  Change from Baseline at Week 24 | -2.9 (3.25) | -2.6 (3.06) | -2.9 (2.45) | -1.9 (2.69)
  Change from Baseline at Week 28: number analyzed (Participants) | 3 | 6 | 3 | 1
  Change from Baseline at Week 28 | -2.5 (2.37) | -4.4 (3.65) | -2.0 (2.62) | -4.0 (NA) — SD cannot be calculated for 1 participant
  Change from Baseline at Week 36: number analyzed (Participants) | 4 | 5 | 4 | 1
  Change from Baseline at Week 36 | -2.3 (2.34) | -1.0 (4.68) | -2.4 (2.30) | -3.8 (NA) — SD cannot be calculated for 1 participant
  Change from Baseline at Week 48: number analyzed (Participants) | 4 | 5 | 4 | 1
  Change from Baseline at Week 48 | -1.7 (1.54) | -2.0 (3.77) | -1.8 (1.41) | -2.6 (NA) — SD cannot be calculated for 1 participant

56. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 50% Improvement (PASI50) Response at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI50, the improvement threshold from baseline in PASI score is 50%. A higher score indicates more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 16 | 17 | 16
percentage of participants
  Week 4: number analyzed (Participants) | 15 | 17 | 15
  Week 4 | 13.3 [0.0 to 33.9] | 35.3 [9.6 to 61.0] | 13.3 [0.0 to 33.9]
  Week 8: number analyzed (Participants) | 15 | 17 | 14
  Week 8 | 40.0 [11.9 to 68.1] | 41.2 [14.8 to 67.5] | 35.7 [7.0 to 64.4]
  Week 12: number analyzed (Participants) | 15 | 17 | 14
  Week 12 | 60.0 [31.9 to 88.1] | 29.4 [4.8 to 54.0] | 42.9 [13.4 to 72.4]
  Week 16: number analyzed (Participants) | 14 | 17 | 14
  Week 16 | 64.3 [35.6 to 93.0] | 35.3 [9.6 to 61.0] | 35.7 [7.0 to 64.4]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-31.0 to 31.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 22.0, 95% CI 2-sided [-12.8 to 56.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 4.3, 95% CI 2-sided [-37.9 to 46.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 5.5, 95% CI 2-sided [-35.4 to 46.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 17.1, 95% CI 2-sided [-25.6 to 59.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = -13.4, 95% CI 2-sided [-53.7 to 26.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 28.6, 95% CI 2-sided [-14.1 to 71.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = -0.4, 95% CI 2-sided [-40.8 to 39.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

57. Secondary Outcome: Percentage of Participants Who Achieved PASI50 Response at Weeks 20, 24, 28, 36, and 48 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: as for outcome 56
Time Frame: Weeks 20, 24, 28, 36, and 48
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 16 | 17 | 5 | 2
percentage of participants
  Week 20: number analyzed (Participants) | 7 | 7 | 5 | 2
  Week 20 | 57.1 [13.3 to 100.0] | 57.1 [13.3 to 100.0] | 40.0 [0.0 to 92.9] | 0 [0.0 to 25.0]
  Week 24: number analyzed (Participants) | 6 | 7 | 4 | 2
  Week 24 | 83.3 [45.2 to 100.0] | 57.1 [13.3 to 100.0] | 75.0 [20.1 to 100.0] | 50.0 [0.0 to 100.0]
  Week 28: number analyzed (Participants) | 2 | 6 | 3 | 1
  Week 28 | 100.0 [75.0 to 100.0] | 66.7 [20.6 to 100.0] | 66.7 [0.0 to 100.0] | 100.0 [50.0 to 100.0]
  Week 36: number analyzed (Participants) | 3 | 5 | 4 | 1
  Week 36 | 66.7 [0.0 to 100.0] | 60.0 [7.1 to 100.0] | 75.0 [20.1 to 100.0] | 100.0 [50.0 to 100.0]
  Week 48: number analyzed (Participants) | 3 | 5 | 4 | 1
  Week 48 | 66.7 [0.0 to 100.0] | 60.0 [7.1 to 100.0] | 50.0 [0.0 to 100.0] | 0 [0.0 to 50.0]

58. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 75% Improvement (PASI75) Response at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI75, the improvement threshold from baseline in PASI score is 75%. A higher score indicates more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 16 | 17 | 16
percentage of participants
  Week 4: number analyzed (Participants) | 15 | 17 | 15
  Week 4 | 13.3 [0.0 to 33.9] | 17.6 [0.0 to 38.7] | 6.7 [0.0 to 22.6]
  Week 8: number analyzed (Participants) | 15 | 17 | 14
  Week 8 | 13.3 [0.0 to 33.9] | 17.6 [0.0 to 38.7] | 7.1 [0.0 to 24.2]
  Week 12: number analyzed (Participants) | 15 | 17 | 14
  Week 12 | 40.0 [11.9 to 68.1] | 17.6 [0.0 to 38.7] | 21.4 [0.0 to 46.5]
  Week 16: number analyzed (Participants) | 14 | 17 | 14
  Week 16 | 42.9 [13.4 to 72.4] | 23.5 [0.4 to 46.6] | 21.4 [0.0 to 46.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.55, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 6.7, 95% CI 2-sided [-21.3 to 34.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.24, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 11.0, 95% CI 2-sided [-17.4 to 39.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.47, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 6.2, 95% CI 2-sided [-22.6 to 35.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.25, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 10.5, 95% CI 2-sided [-18.6 to 39.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.44, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 18.6, 95% CI 2-sided [-21.1 to 58.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.68, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = -3.8, 95% CI 2-sided [-38.4 to 30.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.33, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 21.4, 95% CI 2-sided [-19.4 to 62.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.98, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Difference in response rates = 2.1, 95% CI 2-sided [-33.9 to 38.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

59. Secondary Outcome: Percentage of Participants Who Achieved PASI75 Response at Weeks 20, 24, 28, 36, and 48 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: as for outcome 58
Time Frame: Weeks 20, 24, 28, 36, and 48
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 16 | 17 | 5 | 2
percentage of participants
  Week 20: number analyzed (Participants) | 7 | 7 | 5 | 2
  Week 20 | 14.3 [0.0 to 47.4] | 42.9 [0.0 to 86.7] | 0 [0.0 to 10.0] | 0 [0.0 to 25.0]
  Week 24: number analyzed (Participants) | 6 | 7 | 4 | 2
  Week 24 | 50.0 [1.7 to 98.3] | 42.9 [0.0 to 86.7] | 75.0 [20.1 to 100.0] | 0 [0.0 to 25.0]
  Week 28: number analyzed (Participants) | 2 | 6 | 3 | 1
  Week 28 | 0 [0.0 to 25.0] | 50.0 [1.7 to 98.3] | 66.7 [0.0 to 100.0] | 0 [0.0 to 50.0]
  Week 36: number analyzed (Participants) | 3 | 5 | 4 | 1
  Week 36 | 66.7 [0.0 to 100.0] | 40.0 [0.0 to 92.9] | 50.0 [0.0 to 100.0] | 0 [0.0 to 50.0]
  Week 48: number analyzed (Participants) | 3 | 5 | 4 | 1
  Week 48 | 0 [0.0 to 16.7] | 20.0 [0.0 to 65.1] | 25.0 [0.0 to 79.9] | 0 [0.0 to 50.0]

60. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 90% Improvement (PASI90) Response at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI90, the improvement threshold from baseline in PASI score is 90%. A higher score indicates more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 16 | 17 | 16
percentage of participants
  Week 4: number analyzed (Participants) | 15 | 17 | 15
  Week 4 | 6.7 [0.0 to 22.6] | 5.9 [0.0 to 20.0] | 6.7 [0.0 to 22.6]
  Week 8: number analyzed (Participants) | 15 | 17 | 14
  Week 8 | 13.3 [0.0 to 33.9] | 5.9 [0.0 to 20.0] | 0 [0.0 to 3.6]
  Week 12: number analyzed (Participants) | 15 | 17 | 14
  Week 12 | 6.7 [0.0 to 22.6] | 5.9 [0.0 to 20.0] | 21.4 [0.0 to 46.5]
  Week 16: number analyzed (Participants) | 14 | 17 | 14
  Week 16 | 28.6 [1.3 to 55.8] | 11.8 [0.0 to 30.0] | 7.1 [0.0 to 24.2]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-24.5 to 24.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = -0.8, 95% CI 2-sided [-23.9 to 22.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 13.3, 95% CI 2-sided [-10.8 to 37.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 5.9, 95% CI 2-sided [-11.8 to 23.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = -14.8, 95% CI 2-sided [-46.6 to 17.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = -15.5, 95% CI 2-sided [-46.3 to 15.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 21.4, 95% CI 2-sided [-13.0 to 55.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 4.6, 95% CI 2-sided [-22.3 to 31.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

61. Secondary Outcome: Percentage of Participants Who Achieved PASI90 Response at Weeks 20, 24, 28, 36, and 48 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: as for outcome 60
Time Frame: Weeks 20, 24, 28, 36, and 48
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Filgotinib 100 mg From Placebo (LTE): Filgotinib 100 mg tablet orally once daily+ PTM filgotinib 200 mg tablet orally once daily or up to 44 weeks. Participants received placebo in the Main Study.
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 16 | 17 | 5 | 2
percentage of participants
  Week 20: number analyzed (Participants) | 7 | 7 | 5 | 2
  Week 20 | 0 [0.0 to 7.1] | 14.3 [0.0 to 47.4] | 0 [0.0 to 10.0] | 0 [0.0 to 25.0]
  Week 24: number analyzed (Participants) | 6 | 7 | 4 | 2
  Week 24 | 33.3 [0.0 to 79.4] | 14.3 [0.0 to 47.4] | 0 [0.0 to 12.5] | 0 [0.0 to 25.0]
  Week 28: number analyzed (Participants) | 2 | 6 | 3 | 1
  Week 28 | 0 [0.0 to 25.0] | 16.7 [0.0 to 54.8] | 0 [0.0 to 16.7] | 0 [0.0 to 50.0]
  Week 36: number analyzed (Participants) | 3 | 5 | 4 | 1
  Week 36 | 0 [0.0 to 16.7] | 0 [0.0 to 10.0] | 0 [0.0 to 12.5] | 0 [0.0 to 50.0]
  Week 48: number analyzed (Participants) | 3 | 5 | 4 | 1
  Week 48 | 0 [0.0 to 16.7] | 0 [0.0 to 10.0] | 25.0 [0.0 to 79.9] | 0 [0.0 to 50.0]

62. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 100% Improvement (PASI100) Response at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI100, the improvement threshold from baseline in PASI score is 100%. A higher score indicates more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 16 | 17 | 16
percentage of participants
  Week 4: number analyzed (Participants) | 15 | 17 | 15
  Week 4 | 0 [0.0 to 3.3] | 5.9 [0.0 to 20.0] | 0 [0.0 to 3.3]
  Week 8: number analyzed (Participants) | 15 | 17 | 14
  Week 8 | 6.7 [0.0 to 22.6] | 5.9 [0.0 to 20.0] | 0 [0.0 to 3.6]
  Week 12: number analyzed (Participants) | 15 | 17 | 14
  Week 12 | 0 [0.0 to 3.3] | 5.9 [0.0 to 20.0] | 0 [0.0 to 3.6]
  Week 16: number analyzed (Participants) | 14 | 17 | 14
  Week 16 | 0 [0.0 to 3.6] | 5.9 [0.0 to 20.0] | 0 [0.0 to 3.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-6.7 to 6.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 5.9, 95% CI 2-sided [-11.6 to 23.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 6.7, 95% CI 2-sided [-12.9 to 26.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 5.9, 95% CI 2-sided [-11.8 to 23.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-6.9 to 6.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 5.9, 95% CI 2-sided [-11.8 to 23.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-7.1 to 7.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 5.9, 95% CI 2-sided [-11.8 to 23.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

63. Secondary Outcome: Percentage of Participants Who Achieved PASI100 Response at Weeks 20, 24, 28, 36, and 48 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: as for outcome 62
Time Frame: Weeks 20, 24, 28, 36, and 48
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 16 | 17 | 5 | 2
percentage of participants
  Week 20: number analyzed (Participants) | 7 | 7 | 5 | 2
  Week 20 | 0 [0.0 to 7.1] | 14.3 [0.0 to 47.4] | 0 [0.0 to 10.0] | 0 [0.0 to 25.0]
  Week 24: number analyzed (Participants) | 6 | 7 | 4 | 2
  Week 24 | 0 [0.0 to 8.3] | 14.3 [0.0 to 47.4] | 0 [0.0 to 12.5] | 0 [0.0 to 25.0]
  Week 28: number analyzed (Participants) | 2 | 6 | 3 | 1
  Week 28 | 0 [0.0 to 25.0] | 16.7 [0.0 to 54.8] | 0 [0.0 to 16.7] | 0 [0.0 to 50.0]
  Week 36: number analyzed (Participants) | 3 | 5 | 4 | 1
  Week 36 | 0 [0.0 to 16.7] | 0 [0.0 to 10.0] | 0 [0.0 to 12.5] | 0 [0.0 to 50.0]
  Week 48: number analyzed (Participants) | 3 | 5 | 4 | 1
  Week 48 | 0 [0.0 to 16.7] | 0 [0.0 to 10.0] | 25.0 [0.0 to 79.9] | 0 [0.0 to 50.0]

64. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index at Weeks 4, 8, 12, and 16 in Participants With Enthesitis at Baseline
Description: The enthesitis examination is based on the 16 anatomical sites: the medial epicondyle (left and right), the lateral epicondyle (left and right), the supraspinatus insertion (left and right), the bilateral greater trochanter (left and right), the quadriceps tendon insertion into superior border of patella (left and right), the patellar ligament insertion into inferior pole of patella or tibial tuberosity (left and right), the achilles tendon insertion (left and right), and the plantar fascia insertion (left and right). Enthesitis at each site is scored as either 0 (enthesitis absent) and 1 (enthesitis present). SPARCC enthesitis index has an overall total score ranging from 0 to 16. Higher score indicates a greater number of sites that are affected by enthesitis. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with enthesitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 22 | 22 | 24
score on a scale
  Change from Baseline at Week 4 | -2 (3.8) | -2 (2.3) | 0 (2.7)
  Change from Baseline at Week 8: number analyzed (Participants) | 20 | 22 | 24
  Change from Baseline at Week 8 | -2 (4.9) | -2 (3.2) | -1 (1.9)
  Change from Baseline at Week 12: number analyzed (Participants) | 20 | 22 | 24
  Change from Baseline at Week 12 | -2 (5.1) | -3 (3.2) | -1 (2.8)
  Change from Baseline at Week 16: number analyzed (Participants) | 19 | 21 | 24
  Change from Baseline at Week 16 | -2 (5.6) | -3 (2.9) | -2 (2.2)

65. Secondary Outcome: Change From Baseline in SPARCC Enthesitis Index at Weeks 20, 24, 28, 36, and 48 in Participants With Enthesitis at Baseline
Description: as for outcome 64
Time Frame: Baseline, 20, 24, 28, 36, and 48 weeks
Population: Participants in the FAS with enthesitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 9 | 5
score on a scale
  Change from Baseline at Week 20: number analyzed (Participants) | 10 | 13 | 9 | 5
  Change from Baseline at Week 20 | -3 (5.2) | -4 (3.6) | 0 (2.4) | 0 (1.1)
  Change from Baseline at Week 24: number analyzed (Participants) | 11 | 11 | 7 | 5
  Change from Baseline at Week 24 | -3 (5.3) | -3 (4.3) | 0 (0.4) | -1 (0.8)
  Change from Baseline at Week 28: number analyzed (Participants) | 6 | 7 | 4 | 4
  Change from Baseline at Week 28 | -3 (6.9) | -5 (5.4) | 0 (1.7) | 0 (0.8)
  Change from Baseline at Week 36: number analyzed (Participants) | 7 | 7 | 4 | 4
  Change from Baseline at Week 36 | -4 (5.3) | -5 (5.3) | 0 (2.1) | 1 (1.7)
  Change from Baseline at Week 48: number analyzed (Participants) | 6 | 6 | 4 | 4
  Change from Baseline at Week 48 | -6 (5.3) | -6 (5.8) | -1 (1.0) | 0 (2.0)

66. Secondary Outcome: Change From Baseline in Leeds Dactylitis Index (LDI) at Weeks 4, 8, 12, and 16 in Participants With Dactylitis at Baseline
Description: LDI quantitatively measures dactylitis using the circumference of involved digits and control digits and tenderness of involved digits. Digits affected by dactylitis are defined as those with an at least 10% difference in the ratio of circumference of the affected digit to the contralateral digit. The control digit is either the contralateral digit (digit on opposite hand or foot), or if the contralateral digit is also affected, values from a standard reference table. LDI measures the ratio of the circumference of affected digit to circumference of digit on contralateral hand or foot using a Leeds Dactylometer. LDI score is calculated based on circumference of the dactylitic finger/toe (mm), circumference of the contralateral digit (mm), tenderness score (0 = no tenderness, 1 = tender). Tenderness of affected digits is assessed on a scale from 0 (no tenderness) to 3 (tender and withdrawn). A higher LDI indicates worse dactylitis. Negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with dactylitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 15 | 6 | 9
score on a scale
  Change from Baseline at Week 4 | -18.8 (48.27) | -5.3 (15.36) | 13.1 (70.34)
  Change from Baseline at Week 8 | -45.4 (88.15) | -14.4 (26.14) | 23.3 (129.90)
  Change from Baseline at Week 12 | -49.8 (85.77) | -11.8 (11.82) | -15.8 (15.82)
  Change from Baseline at Week 16: number analyzed (Participants) | 14 | 6 | 9
  Change from Baseline at Week 16 | -42.1 (95.15) | -11.7 (6.30) | -16.2 (15.04)

67. Secondary Outcome: Change From Baseline in LDI at Weeks 20, 24, 28, 36, and 48 in Participants With Dactylitis at Baseline
Description: LDI quantitatively measures dactylitis using the circumference of involved digits and control digits and tenderness of involved digits. Digits affected by dactylitis are defined as those with an at least 10% difference in the ratio of circumference of the affected digit to the contralateral digit. The control digit is either the contralateral digit (digit on opposite hand or foot), or if the contralateral digit is also affected, values from a standard reference table. LDI measures the ratio of the circumference of affected digit to circumference of digit on contralateral hand or foot using a Leeds Dactylometer. LDI score is calculated based on the circumference of the dactylitic finger/toe (mm), circumference of contralateral digit (mm), tenderness score (0 = no tenderness, 1 = tender). Tenderness of affected digits is assessed on a scale from 0 (no tenderness) to 3 (tender and withdrawn). A higher LDI indicates worse dactylitis. Negative change from baseline indicates improvement.
Time Frame: Baseline, 20, 24, 28, 36, and 48 weeks
Population: Participants in the FAS with dactylitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 15 | 6 | 4 | 2
score on a scale
  Change from Baseline at Week 20: number analyzed (Participants) | 7 | 4 | 4 | 2
  Change from Baseline at Week 20 | -79.5 (120.99) | -9.7 (6.78) | 0.0 (0.00) | 0.0 (0.00)
  Change from Baseline at Week 24: number analyzed (Participants) | 6 | 3 | 2 | 2
  Change from Baseline at Week 24 | -94.2 (125.41) | -13.0 (2.37) | 0.0 (0.00) | 0.0 (0.00)
  Change from Baseline at Week 28: number analyzed (Participants) | 3 | 2 | 2 | 1
  Change from Baseline at Week 28 | -164.6 (147.22) | -11.8 (1.64) | 0.0 (0.00) | 0.0 (NA) — SD cannot be calculated for 1 participant.
  Change from Baseline at Week 36: number analyzed (Participants) | 4 | 2 | 1 | 1
  Change from Baseline at Week 36 | -123.4 (145.68) | -11.8 (1.64) | 0.0 (NA) — SD cannot be calculated for 1 participant. | 0.0 (NA) — SD cannot be calculated for 1 participant.
  Change from Baseline at Week 48: number analyzed (Participants) | 4 | 2 | 1 | 1
  Change from Baseline at Week 48 | -123.4 (145.68) | -11.8 (1.64) | 0.0 (NA) — SD cannot be calculated for 1 participant. | 0.0 (NA) — SD cannot be calculated for 1 participant.

68. Secondary Outcome: Change From Baseline in Tender Dactylitis Count (TDC) at Weeks 4, 8, 12, and 16 in Participants With Dactylitis at Baseline
Description: Tender score (0 = no tenderness, 1 = tender, 2 = tender and wince, 3 = tender and withdraw) is collected for Dactylitis Assessments on the Dactylitis Score Sheet that is used for calculation of LDI total score. Tender dactylitis count (TDC) equals the number of tender fingers and toes (tendor score >0). For participants with dactylitis status absent for all the fingers and toes, the TDC is set as 0. The total score range of TDC is from 0 to 60, higher scores indicate greater presence of dactylitis. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with dactylitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender dactylitis count
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 15 | 6 | 9
tender dactylitis count
  Change from Baseline at Week 4 | -1 (2.2) | 1 (2.7) | 0 (3.1)
  Change from Baseline at Week 8 | -3 (5.1) | 1 (3.7) | 1 (7.1)
  Change from Baseline at Week 12 | -3 (5.1) | -1 (0.8) | -1 (1.0)
  Change from Baseline at Week 16: number analyzed (Participants) | 14 | 6 | 9
  Change from Baseline at Week 16 | -3 (5.3) | -1 (0.5) | -1 (0.8)

69. Secondary Outcome: Change From Baseline in TDC at Weeks 20, 24, 28, 36, and 48 in Participants With Dactylitis at Baseline
Description: as for outcome 68
Time Frame: Baseline, 20, 24, 28, 36, and 48 weeks
Population: Participants in the FAS with dactylitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender dactylitis count
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 15 | 6 | 4 | 2
tender dactylitis count
  Change from Baseline at Week 20: number analyzed (Participants) | 7 | 4 | 4 | 2
  Change from Baseline at Week 20 | -5 (7.2) | -1 (0.5) | 0 (0.0) | 0 (0.0)
  Change from Baseline at Week 24: number analyzed (Participants) | 6 | 3 | 2 | 2
  Change from Baseline at Week 24 | -6 (7.4) | -1 (0.0) | 0 (0.0) | 0 (0.0)
  Change from Baseline at Week 28: number analyzed (Participants) | 3 | 2 | 2 | 1
  Change from Baseline at Week 28 | -10 (9.0) | -1 (0.0) | 0 (0.0) | 0 (NA) — SD cannot be calculated for 1 participant.
  Change from Baseline at Week 36: number analyzed (Participants) | 4 | 2 | 1 | 1
  Change from Baseline at Week 36 | -7 (8.8) | -1 (0.0) | 0 (NA) — SD cannot be calculated for 1 participant. | 0 (NA) — SD cannot be calculated for 1 participant.
  Change from Baseline at Week 48: number analyzed (Participants) | 4 | 2 | 1 | 1
  Change from Baseline at Week 48 | -7 (8.8) | -1 (0.0) | 0 (NA) — SD cannot be calculated for 1 participant. | 0 (NA) — SD cannot be calculated for 1 participant.

70. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Weeks 2, 4, 8, 12, and 16
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). When 6 or more categories are non-missing, total possible score is 3. If more than 2 categories are missing, the HAQ-DI score is set to missing. A negative change from baseline indicates improvement (less disability).
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 34 | 33 | 36
  Change from Baseline at Week 2 | -0.13 (0.343) | -0.04 (0.277) | -0.03 (0.228)
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | -0.16 (0.320) | -0.06 (0.364) | -0.07 (0.273)
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 34 | 34
  Change from Baseline at Week 8 | -0.29 (0.412) | -0.07 (0.471) | -0.10 (0.337)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 34 | 34
  Change from Baseline at Week 12 | -0.38 (0.506) | -0.15 (0.401) | -0.14 (0.342)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 33
  Change from Baseline at Week 16 | -0.38 (0.489) | -0.09 (0.456) | -0.08 (0.328)
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.19, MMRM — P-value was provided from MMRM including treatment, visit (categorical), treatment by visit, stratification factors, baseline value as fixed effects, participants being the random effect; LS Mean Treatment Difference = -0.09, 95% CI 2-sided [-0.22 to 0.04], Standard Error of Mean 0.066
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.84, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = -0.01, 95% CI 2-sided [-0.15 to 0.12], Standard Error of Mean 0.067
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.30, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = -0.08, 95% CI 2-sided [-0.22 to 0.07], Standard Error of Mean 0.073
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.89, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 0.01, 95% CI 2-sided [-0.14 to 0.16], Standard Error of Mean 0.074
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.064, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = -0.18, 95% CI 2-sided [-0.37 to 0.01], Standard Error of Mean 0.096
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.88, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 0.01, 95% CI 2-sided [-0.17 to 0.20], Standard Error of Mean 0.096
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.023, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = -0.23, 95% CI 2-sided [-0.43 to -0.03], Standard Error of Mean 0.099
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.75, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = -0.03, 95% CI 2-sided [-0.23 to 0.17], Standard Error of Mean 0.099
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.005, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = -0.31, 95% CI 2-sided [-0.51 to -0.10], Standard Error of Mean 0.106
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.54, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = -0.07, 95% CI 2-sided [-0.27 to 0.14], Standard Error of Mean 0.105

71. Secondary Outcome: Change From Baseline in HAQ-DI Score at Weeks 18, 20, 24, 28, 36, 48, and 60
Description: as for outcome 70
Time Frame: Baseline, 18, 20, 24, 28, 36, 48, and 60 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 18 | 20 | 10 | 8
score on a scale
  Change from Baseline at Week 18: number analyzed (Participants) | 15 | 18 | 8 | 8
  Change from Baseline at Week 18 | -0.42 (0.403) | -0.09 (0.481) | -0.11 (0.254) | -0.02 (0.156)
  Change from Baseline at Week 20: number analyzed (Participants) | 13 | 19 | 10 | 8
  Change from Baseline at Week 20 | -0.38 (0.468) | -0.14 (0.573) | -0.28 (0.558) | -0.02 (0.356)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 16 | 7 | 7
  Change from Baseline at Week 24 | -0.21 (0.431) | -0.30 (0.546) | -0.29 (0.672) | -0.11 (0.168)
  Change from Baseline at Week 28: number analyzed (Participants) | 8 | 11 | 4 | 5
  Change from Baseline at Week 28 | -0.23 (0.430) | -0.33 (0.485) | -0.63 (0.685) | -0.13 (0.234)
  Change from Baseline at Week 36: number analyzed (Participants) | 9 | 10 | 4 | 5
  Change from Baseline at Week 36 | -0.36 (0.345) | -0.29 (0.417) | -0.25 (0.777) | -0.20 (0.259)
  Change from Baseline at Week 48: number analyzed (Participants) | 8 | 9 | 4 | 3
  Change from Baseline at Week 48 | -0.41 (0.346) | -0.25 (0.428) | -0.44 (0.725) | -0.04 (0.191)
  Change from Baseline at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 2
  Change from Baseline at Week 60 | 0.00 (NA) — SD cannot be calculated for 1 participant. | -0.25 (NA) — SD cannot be calculated for 1 participant. | -0.38 (0.000) | -0.19 (0.265)

72. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) Score at Weeks 4 and 16
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 0 to 52. Higher scores indicate less fatigue. Positive change in value indicates improvement (no or less severity of fatigue).
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | 4.8 (6.80) | 2.3 (5.94) | 2.5 (8.23)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 34
  Change from Baseline at Week 16 | 6.9 (11.56) | 1.9 (7.93) | 0.6 (11.14)
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.43, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 1.3, 95% CI 2-sided [-1.9 to 4.5], Standard Error of Mean 1.64
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.81, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = -0.4, 95% CI 2-sided [-3.6 to 2.9], Standard Error of Mean 1.64
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.040, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 5.1, 95% CI 2-sided [0.2 to 9.9], Standard Error of Mean 2.43
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.58, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 1.4, 95% CI 2-sided [-3.4 to 6.1], Standard Error of Mean 2.41

73. Secondary Outcome: Change From Baseline in FACIT-Fatigue Scale Score at Week 48
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 0 to 52. Higher scores indicate better quality of life. Positive change in value indicates improvement (no or less severity of fatigue).
Time Frame: Baseline, Week 48
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 17 | 19 | 10 | 8
score on a scale | 6.9 (11.27) | 4.4 (11.76) | 5.1 (9.09) | 3.0 (7.63)

74. Secondary Outcome: Change From Baseline in Mental Component Score (MCS) of the 36-Item Short-Form Version 2 (SF-36v2) at Weeks 4 and 16
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (MCS and PCS). MCS consists of social functioning, vitality, mental health, and role-emotional scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning. A positive change from baseline indicated improvement (better health status).
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | 1.4 (7.91) | 1.0 (5.07) | -0.2 (8.48)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 34
  Change from Baseline at Week 16 | 3.3 (9.84) | 1.8 (8.12) | 0.7 (9.43)

75. Secondary Outcome: Change From Baseline in MCS of the SF-36v2 at Week 48
Description: as for outcome 74
Time Frame: Baseline, Week 48
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 17 | 19 | 10 | 8
score on a scale | 2.3 (10.55) | 1.5 (8.74) | -0.5 (4.13) | -1.4 (7.51)

76. Secondary Outcome: Change From Baseline in Physical Component Score (PCS) of the SF-36v2 at Weeks 4 and 16
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (MCS and PCS). PCS consists of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning. A positive change from baseline indicates improvement (better health status).
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 36 | 34 | 36
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 36 | 34 | 35
  Change from Baseline at Week 4 | 2.1 (4.95) | 2.2 (3.92) | 0.8 (5.61)
  Change from Baseline at Week 16: number analyzed (Participants) | 32 | 33 | 34
  Change from Baseline at Week 16 | 4.6 (6.43) | 2.6 (5.80) | 0.6 (5.95)
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.40, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 0.9, 95% CI 2-sided [-1.2 to 3.1], Standard Error of Mean 1.09
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.28, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 1.2, 95% CI 2-sided [-1.0 to 3.4], Standard Error of Mean 1.10
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.011, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 3.8, 95% CI 2-sided [0.9 to 6.7], Standard Error of Mean 1.46
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.14, MMRM — [p-value comment as in outcome 70, analysis 1]; LS Mean Treatment Difference = 2.1, 95% CI 2-sided [-0.7 to 5.0], Standard Error of Mean 1.45

77. Secondary Outcome: Change From Baseline in PCS of the SF-36v2 at Week 48
Description: as for outcome 76
Time Frame: Baseline, Week 48
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Number analyzed (Participants) | 17 | 19 | 10 | 8
score on a scale | 1.7 (7.27) | 3.2 (7.54) | 3.8 (8.51) | -1.9 (4.74)

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 63 weeks plus 30 days; All-Cause Mortality: Randomization up to 63 weeks plus 30 days
Description: Adverse Events: Safety Analysis Set included all participants who took at least 1 dose of study drug. All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study.
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Placebo (Main Study) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34 | 0/36 | 0/18 | 0/20 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/34 | 0/36 | 1/18 | 1/20 | 0/10 | 2/8
Other Adverse Events (participants affected / at risk) | 7/36 | 4/34 | 9/36 | 10/18 | 7/20 | 5/10 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (Main Study) (N=36) | Filgotinib 100 mg (Main Study) (N=34) | Placebo (Main Study) (N=36) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) (N=18) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) (N=20) | Filgotinib 200 mg From Placebo (LTE) (N=10) | Filgotinib 100 mg From Placebo (LTE) (N=8)
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (Main Study) (N=36) | Filgotinib 100 mg (Main Study) (N=34) | Placebo (Main Study) (N=36) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) (N=18) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) (N=20) | Filgotinib 200 mg From Placebo (LTE) (N=10) | Filgotinib 100 mg From Placebo (LTE) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular myasthenia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 2 | 1 | 1 | 1 | 2
Ear infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure systolic increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mechanical acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT04115839/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT04115839/SAP_001.pdf